

**Protocol Number:** AVXS-101-CL-101 (formerly AVXS-101)

**IND Number:** 15699

**Protocol Title:** Phase I Gene Transfer Clinical Trial for Spinal

Muscular Atrophy Type 1 Delivering AVXS-101

**Indication Studied:** Spinal muscular atrophy Type 1

**Sponsor Address:** 2275 Half Day Road, Suite 160

Bannockburn, IL 60015

**Protocol Version/Date:** Version 14.0 / 21 April 2016

The study will be completed according to the guidelines of Good Clinical Practice. Compliance with this standard provides public assurance that the rights, safety, and well-being of trial subjects are protected, consistent with the principles that have their origin in the Declaration of Helsinki.

# **Confidentiality Statement**

The information in this document contains trade and commercial information that is privileged or confidential and may not be disclosed unless such disclosure is required by federal or state law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you which is indicated as privileged or confidential.

# 1 ADMINISTRATIVE INFORMATION

# 1.1 Summary of Changes

This version of the protocol reflects the change in sponsorship of the study from Sophia's Cure and NCH to AveXis, Inc. This protocol was prepared utilizing the AveXis, Inc. clinical study protocol template, and combines the latest version of the protocol, version 13.0 dated 10 June 2015 and the Protocol Addendum #2 version 1.0 dated 24 June 2015.

The following table outlines the transfer of protocol sections from the previous NCH version(s) of the protocol template to the current AveXis, Inc. protocol template.

 Table 1
 Summary of Protocol Section Changes and Additions

| | NCH | | AveXis |
|---|---|---|---|
| Section # | Section Title | Section # | Section Title |
| | Sections Existing in previous versions of protocol(s) | | |
| 1.0 | Synopsis | 2.0 | Synopsis |
| 2.0 | Abstract | 5 | Introduction |
| 3.0 | Clinical Trial and Principal Investigator | N/A | N/A |
| 3.2 | Rationale for Gene Transfer to SMA Type 1 Patients | 5.2 | Rationale for Gene Transfer to SMA Type 1 Patients |
| 3.3 | Background and Preliminary Data | 5.1 | Background and Preliminary Data |
| 4.0 | Preliminary Data | 5.3 | Non-clinical Studies |
| 5.0 | Research | 6 | Trial Objectives and Purpose |
| 5.2 | Pre-Treatment Assessment | 8 | Selection and Withdrawal of Subjects |
| 5.3 | Dosing Plan | 9, 10.5, 10.6 | Treatment of Subjects, Administration, Dose Escalation |
| 5.4 | Clinical Trial Monitoring Plan | 11 | Assessments |
| 5.5 | Outcome Measures | 6 (6.1–6.3) | Trial Objectives and Purpose |
| 5.6 | Statistical Analysis | 13 | Statistics |
| 5.7 | Timeline of Assessments | Table 6 | Schedule of Assessments |
| 6.0 | Dose Limiting Toxicity | 11.1.1 | Dose Limiting Toxicity |
| 6.1 | The classification for adverse events | 11.1.1 | Dose Limiting Toxicity |
| 6.3 | Stopping/Discontinuation Rules | 8.3 | Subject Withdrawal Criteria |
| 6.4 | Dose Escalation | 10.6 | Dose Escalation |
| 7.0 | Adverse Event Monitoring and Reporting | 12 | Adverse and Serious Adverse Events,<br>Relationship to Study Drug, Recording<br>Adverse Events, Reporting Adverse<br>Events |
| 8.0 | Study Reports | N/A | N/A |
| | | | Study reports are a sponsor responsibility, outlined in sponsor SOPs |
| 8.3 | Data Safety Monitoring Plan | 13 | Data Safety Monitoring Board |
| 8.4 | Clinical Monitoring of the Study | 15.1 | Study Monitoring |
| 9.0 | References | 19 | References |

| NCH | | AveXis | |
|---|---|---|---|
| Section # | Section Title | Section # | Section Title |
| Addendum 1 | Autopsy Plan | Appendix 2 | Autopsy Plan |
| | New Sections that were not present | in previous ver | rsion(s) of protocol(s) |
| N/A | N/A | 15.2 | Audits and Inspections |
| N/A | N/A | 16 | Ethics |
| N/A | N/A | 17 | Data Handling and Recordkeeping |
| N/A | N/A | 18 | Publication Policy |
| | N/A | Appendix 1 | Declaration of Helsinki |
| | N/A | Appendix 3 | CHOP-INTEND |
| | N/A | Appendix 4 | Bayley Scale of Infant Development, version 3 |
| | N/A | Appendix 5 | Gross Motor Skills Checklist |
| ŗ | The following sections were overhauled to | | - · |
| | supporting AveXis, Inc | , as managing | sponsor |
| N/A | N/A | 12 | Adverse and Serious Adverse Events |
| N/A | N/A | 13 | Data Safety Monitoring Board |

The section below highlights content changes represented in this version of the protocol. Language deleted from the previous version of the protocol appears in *italics*. Language added to the previous version of the protocol appears in **bold**.

# Section 6.2: Secondary Objectives

A secondary outcome will include time from birth to either (a) requirement of  $\geq$ 16-hour respiratory assistance per day (includes BiPAP) continuously for >2 weeks in the absence of an acute reversible illness or (b) death.

Secondary outcomes will also include the change in CHOP-INTEND from baseline score and demonstration of improvement of motor function and muscle strength as determined by achievement of significant development milestones including but not limited to the ability to sit alone and roll over unassisted. Additionally, AveXis, Inc. may opt to provide videos of the physical exams, CHOP-INTEND assessments, and/or Bayley Scale assessments to an independent, blinded reviewer for confirmation of the development milestones.

## Rationale for Change

Achievement of motor milestones will serve as a more clinically meaningfully efficacy endpoint.

# Section 6.3: Exploratory Objectives

Exploratory outcome measures will be tested during the study as part of the program and product development plan; however if exploratory measurement results show efficacy and primary outcomes do not reach statistical significance, the only interpretation is that the results show a trend toward benefit but can never supersede primary measures. These exploratory outcome measures will include:

 ACTIVE-mini (Ability Captured Through Interactive Video Evaluation-mini) evaluation of infant movement ability.

- Patient functional measures using the Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP-INTEND). This test has been studied and validated in infants with spinal muscular atrophy and was found to be reliable in this population.<sup>19</sup>
- Bayley Scales of Infant Development version 3 is a standardized, norm-referenced infant assessment. The gross and fine motor portions of this test will administered if the child reaches or exceeds a score of 60 out of 64 on the CHOP-INTEND.
- Motor neuron function will be assessed via evoked compound motor action potentials (CMAP) and motor unit number estimation (MUNE).
- Pathological status of muscles will be quantified by Electrical Impedance Myography (EIM).
- The age at which significant motor milestones are achieved will be assessed using a standard Motor Milestone Development Survey shown in Table 10 in Section 11.1.10.
- Compelling, demonstrable, documented evidence of efficacy as determined by changes in functional abilities as captured during videotaping sessions during site visits and/or captured by subject/parent/legal guardian at home.

# Rationale for Change

Determination that "compelling evidence" of efficacy may be documented via video-taped physical therapy sessions, showing motor milestone achievement.

# Section 7.1: Overall Study Design

The proposed clinical trial is an open-label, single injection ascending dose study of self-complementary AAV9 carrying the SMN gene under the control of a hybrid CMV enhancer/chicken AVXS-101 delivered one-time through a venous catheter inserted into a peripheral vein (arm, leg, or scalp) of Type 1 spinal muscular atrophy subjects.

The primary analysis for efficacy will be assessed when all patients reach 13.6 months of age (a database lock will be performed at the time point at which all patients reach 13.6 months of age). A follow-up safety analysis will be completed at the time point at which the last patient reaches 24 months post-dose.

# Rationale for Change

In a natural history study of SMA Type 1 survival,<sup>20</sup> the distribution of the age at reaching the combined endpoint of death or respiratory failure differed by SMN2 copy number. The median age at the combined endpoint for subjects with two (2) SMN2 copies was 10.5 (IQR 8.1-13.6). Therefore, 13.6 months is the expected age at which 75% of SMA Type 1 patients with two (2) SMN2 copies will have met the endpoint of death and/or respiratory failure.

The following are procedures that are being conducted for study purposes, but were not described/outlined as appropriate in previous versions of the protocol(s):

# Section 8.1 Inclusion Criteria

Subjects must meet all of the following Inclusion Criteria:

1. Six months of age and younger<sup>1</sup> at day of vector infusion with Type 1 SMA as defined by the following features:

- a. Bi-allelic SMN1 gene mutations (deletion or point mutation) with two copies of SMN2 (no more and no fewer).
- b. Patients 6 months and younger with a disease onset up to 6 months of age
- c. Hypotonia by clinical evaluation with delay in motor skills, poor head control, round shoulder posture and hypermobility of joints.
- First nine subjects enrolled under previous version(s) of the protocol could be nine months of age or younger. Inclusion revised to reflect six months of age or younger in 24 Jun 2015 Protocol Addendum #2.

Initial genetic testing and diagnosis completed at an institution/laboratory other than Nationwide Children's Hospital/Ohio State University is acceptable if proper documentation is received at Nationwide Children's Hospital, verified by the PI, and filed in the patient's medical record.

AveXis, Inc. may opt to confirm all genetic diagnoses through a contracted third-party laboratory utilizing an additional blood sample collected during a post-dose visit.

# Rationale for Change

For clarification purposes, added notation that baseline diagnostic genetic testing was not completed at Nationwide Children's Hospital in all cases. As noted, AveXis, Inc. may opt to have baseline blood samples for all subjects re-tested at a commercial laboratory to ensure consistent results for all subjects in the trial. As these samples would be run after enrollment/dosing was complete, results would not impact subject eligibility.

# Section 11.8.1 CHOP-INTEND

CHOP-INTEND including head control, righting reactions, and trunk movements in supported sitting, supine, and prone positions. Anti-gravity movements in assisted rolling, ventral suspension, and supported standing are also measured. **See Appendix 3.** 

At such time that a subject achieves two consecutive CHOP-INTEND scores of ≥62, a teleconference will be conducted between PI, physical therapist, and AveXis, Inc. to review the subject status and determine whether or not continued CHOP-INTEND assessments are necessary. A decision will be reached and confirmed in writing following the teleconference. If decided that no further assessments are necessary, the physical therapist will cease completion of the CHOP-INTEND assessment at subsequent visits; otherwise CHOP-INTEND assessments will continue monthly.

CHOP-INTEND examinations will be videotaped in accord with the Videotaping Manual.

# Rationale for Change:

As patients on a normal development course age, CHOP-INTEND scores decrease over time as there are portions of the assessment that are specific to infant development. As patients develop out of infancy, they no longer exhibit some motor functions in an appropriate way for some of the assessment sections to be scored. As study subjects achieve a score of 64, more in line with a

normal development course, it would be inappropriate to continue with the CHOP-INTEND for the same reason.

# Section 11.8.2 Bayley Scale of Infant Development version 3

Bayley Scales of Infant Development version 3 is a standardized, norm-referenced infant assessment. The gross and fine motor portions and cognition portions of this test will administered if the child reaches or exceeds a score of 60 out of 64 on the CHOP-INTEND. The gross and fine motor portion will be completed monthly during the first year and the cognition portion will be completed every three months. During the second year all required portions of the Bayley Scale will be conducted every three months, except for subjects still being seen monthly for CHOP-INTEND assessments. For those subjects the gross and fine motor and cognition portions will be administered as in Year 1. See Appendix 4.

Bayley scales examinations will be videotaped in accord with the Videotaping Manual.

# Section 11.9 Development Milestones Checklist

The age at which significant motor milestones are achieved will be assessed using a standard Motor Milestone Development Survey shown in Table 10 and a Gross Motor Skills Checklist shown in Appendix 5. The Gross Motor Skills Checklist was designed by physical therapists at Nationwide Children's Hospital specifically to assess SMA Type 1 subjects in this trial; it is source from a collection of existing motor assessments. See Appendix 5.

Additionally, CHOP-INTEND and Bayley physical therapy assessment videos may be transferred to a centralized reviewer for independent determination of milestones achieved.

## Rationale for Change

The Gross Motor Skills Checklist was developed as an assessment and added to the protocol as a method by which to evaluate subjects achieving a maximum CHOP-INTEND score of 64.

# Section 11.10 Video Evidence

Physical therapy assessments and physician physical examinations required at each study visit will be videotaped in an effort to produce compelling, demonstrable, documented evidence of efficacy as determined by changes in functional abilities. Parent(s)/legal guardian(s) may also share home videos demonstrating achievement of functional abilities. AveXis, Inc. will provide a secure and confidential upload process for transfer and storage of the videos from NCH to a contracted third-party vendor that will compile and arrange videos as per AveXis, Inc. submission requirements. Any/all videos received at AveXis, Inc. or the contracted vendor will be treated as confidential study data and will be the sole property of AveXis, Inc. AveXis, Inc. and the contracted vendor will provide this secure, encrypted transfer and storage solution to properly protect the identities of patients/families on the videos, which may be shared with regulatory agencies and/or the medical community.

Videos will be provided in a blinded fashion to an independent, centralized reviewer for unbiased assessment of milestone achievement.

# Section 11.18 Photographs of Infusion Site

Photographs will be taken of the infusion site at the time points specified in Table 6. AveXis, Inc. will provide a secure and confidential upload process for transfer and storage of the photographs from NCH to a contracted third-party vendor that will compile and arrange photographs as per AveXis, Inc. submission requirements. Any/all photographs received at AveXis, Inc. or the contracted vendor will be treated as confidential study data and will be the sole property of AveXis, Inc. AveXis, Inc. and the contracted vendor will provide this secure, encrypted transfer and storage solution to properly protect the identities of patients/families in the photographs, which may be shared with regulatory agencies and/or the medical community.

# Section 11.19.11 Saliva, Urine, Stool Collection

Saliva, urine, and stool samples will be collected for viral shedding studies. Saliva will be collected from the patient's mouth with a pipette and oral swab.  $200-500~\mu L$  of urine will be collected from patients' soiled diapers by soaking a cotton ball. Pea-sized fecal samples will be collected from patients' soiled diapers. Each of these samples will be placed in a DNAse/RNAse-free Eppendorf tube with locking top. The tubes will be stored in a -80°C freezer.

## Rationale for Change

Saliva, urine, and stool samples will be collected to study viral shedding.

## 1.2 Contact Information

 Table 2
 Important Study Contact Information

| Role in Study | Name | Address and Telephone number |
|---|---|---|
| Clinical Study Leader | Clinical Trials Management -<br>Clinical Operations | 2275 Half Day Road, Suite 160<br>Bannockburn, IL 60015<br>Office: (847) 572-8405 |
| | | Mobile: (773) 818-2111 cwells@avexis.com |
| Responsible Physician | Doug Sproule, MD, AveXis Vice<br>President, Clinical Development | 2275 Half Day Road, Suite 160<br>Bannockburn, IL 60015<br>Office: (847) 572-8406<br>Mobile: (978) 505-2524<br>dsproule@avexis.com |

| Role in Study | Name | Address and Telephone number |
|---|---|---|
| Drug Safety Physician | Gloria Galloway, MD | OSU Safety Monitor |
| NCH Safety Monitor | | Ohio State University |
| | | 395 W 12 <sup>th</sup> Avenue |
| | | Columbus, OH 43210 |
| | | Office: (614) 293-4969 |
| | | Mobile: (614) 937-2417 |
| | | Galloway.58@osu.edu |
| 24-Hour Emergency Contact | Jerry Mendell, MD | NCH |
| | Samiah Al-Zaidy, MD | 700 Children's Drive- WA 3011 |
| | | Columbus, OH 43205 |
| | | Mendell: (614) 355-5247 |
| | | Al-Zaidy: (614) 355-3682 |
| SAE Reporting | AveXis | safetyreporting@avexis.com |
| | | FAX: (847) 510-0775 |
| CRO Project Manager | Toni Miller, Sr. Project Manager, | 1700 Perimeter Park Drive |
| | Novella Clinical | Morrisville, NC 27560, United States |
| | | Office: 919-972-7391 |
| | | Mobile: 765-481-6257 |
| | | tmiller@novellaclinical.com |

Table 3: Study Vendor Listing

| Role in Study | Name | Address |
|---|---|---|
| Clinical Research Organization | Novella | 1700 Perimeter Park Drive<br>Morrisville, NC 27560 |
| Video | Video 1 Productions | 1820 W. Webster Ave., Ste. 201<br>Chicago, IL 60614 |
| Central Laboratory- confirmatory genetic testing | Q <sup>2</sup> Solutions | 200 Forest Street, Suite 200<br>Marlborough, MA 01752 USA |
| Autopsy | Regional Pathology and Autopsy<br>Services, Inc. | Oakland, CA<br>877-330-7727 |

## 2 SYNOPSIS

Name of Sponsor/Company: AveXis, Inc.

Name of Investigational Product: AVXS-101

Name of Active Ingredient: Survival Motor Neuron Gene by Self-Complementary AAV9

Title of Study: Phase I Gene Transfer Clinical Trial for Spinal Muscular Atrophy Type 1 Delivering

AVXS-101

**Study center(s):** Nationwide Children's Hospital

**Principal Investigator:** Jerry Mendell, MD

Studied period (years): Phase of development: 1

Estimated date first patient enrolled: May 2014 Estimated date last patient completed: Jan 2017

# Objectives:

## Primary:

 Determination of safety based on the development of unacceptable toxicity: defined as the occurrence of any one Grade III or higher, unanticipated, treatment-related toxicity.

## Secondary:

• The time from birth until death or until patient requires at least 16-hour per day of ventilation support for breathing for ≥14 consecutive days in the absence of an acute reversible illness, excluding perioperative use.

#### Methodology:

Open-label, dose-escalation clinical trial of AVXS-101 injected intravenously through a peripheral limb vein. Short-term safety will be evaluated over a two year period. Patients will be tested at baseline and return for follow up visits on days 7, 14, 21, 30, followed by once every month through 12 months post dose, and then every three months through two (2) years post infusion. Unscheduled visits may occur if the PI determines that they are necessary.

The primary analysis for efficacy will be assessed when all patients reach 13.6 months of age (a database lock will be performed at the time point at which all patients reach 13.6 months of age). A follow-up safety analysis will be completed at the time point at which the last patient reaches 24 months post-dose.

Upon completion of the 2-year study period, patients will be monitored annually as per standard of care for up to 15 years.

## Number of patients (planned): 15

## Diagnosis and main criteria for inclusion:

## **Inclusion Criteria**

• Six months of age and younger at day of vector infusion with Type 1 SMA as defined by the following features:

- Diagnosis of SMA based on gene mutation analysis with bi-allelic SMN1 mutations (deletion or point mutations) and 2 copies of SMN2.
- Onset of disease at birth: up to 6 months of age.
- Hypotonia by clinical evaluation with delay in motor skills, poor head control, round shoulder posture and hypermobility of joints

#### **Exclusion Criteria**

- Active viral infection (includes HIV or serology positive for hepatitis B or C)
- Use of invasive ventilatory support (tracheotomy with positive pressure) or pulse oximetry <95% saturation at the screening visit.</li>
  - Patients may be managed using non-invasive ventilator support (BiPAP) for less than 16 hours per day at the discretion of their physician or study staff.
- Concomitant illness that in the opinion of the PI creates unnecessary risks for gene transfer
- Concomitant use of any of the following drugs: drugs for treatment of myopathy or neuropathy, agents used to treat diabetes mellitus, or ongoing immunosuppressive therapy or immunosuppressive therapy within 3 months of starting the trial (eg, corticosteroids, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, intravenous immunoglobulin, rituximab)
- Patients with Anti-AAV9 antibody titers >1:50 as determined by ELISA binding immunoassay.
- Abnormal laboratory values considered to be clinically significant (GGT >3 X ULN, Bilirubin ≥3.0 mg/dL, Creatinine ≥1.8 mg/dL, Hgb <8 or >18 g/Dl; WBC >20,000 per cmm)
- Participation in recent SMA treatment clinical trial that in the opinion of the PI creates unnecessary risks for gene transfer.
- Family does not want to disclose patient's study participation with primary care physician and other medical providers.
- Patient with signs of aspiration based on a swallowing test and unwilling to use an alternative method to oral feeding.
- Patients with a single base substitution in SMN2 (c.859G>C in exon 7) will be excluded based on predicted mild phenotype.

## Investigational product, dosage and mode of administration:

Cohort 1 will consist of three (3) SMA patients followed by Cohort 2A with a minimum of three (3) and no more than six (6) SMA patients to receive a single infusion at escalating doses.

- Cohort 1 (Low Dose): 6.7 X 10<sup>13</sup> vg/kg (n=3)
- Cohort 2A (Intermediate Dose):  $2.0 \times 10^{14} \text{ vg/kg}$  ( $n \ge 3$  and  $n \le 6$ )

Cohort 2B and Cohort 3 will each consist of three (3) SMA patients to receive a single infusion at escalating doses.

- Cohort 2B:  $2.0 \times 10^{14} \text{ vg/kg (n=3)}$
- Cohort 3 (High Dose): 3.3 X 10<sup>14</sup> vg/kg (n=3)

Cohort 2B will be done first and if efficacy is favorable but does not fully improve subjects to normal, Cohort 3 at high dose will be implemented.

Treatment of Cohort 3 is permitted based on safety assessment presented in the IND. A score of 8 or higher on the Bayley Scales of Infant Development will be considered the low end of normal.

**Duration of treatment:** The vector will be delivered approximately in 10–20 mL/kg of normal saline infused approximately for 60 minutes.

# Reference therapy, dosage and mode of administration: N/A

## Criteria for evaluation:

## Safety:

• Incidence of Grade III or higher, unanticipated, treatment-related toxicity.

# Efficacy:

- Time to death or until patient requires at least 16-hour per day of ventilation support for breathing for ≥14 consecutive days in the absence of an acute reversible illness, excluding perioperative use
- A successful measure for efficacy for this study will be 50% of SMA Type 1 subjects living independently of 16 or more hours of ventilator support at 2 years.
- Change in CHOP-INTEND from baseline measure score of age.
- To determine efficacy by demonstrating improvement of motor function and muscle strength as determined by achievement of significant development milestones including but not limited to the ability to sit alone and roll over unassisted. Additionally, AveXis, Inc. may opt to provide videos of the physical exams, CHOP-INTEND assessments, and/or Bayley Scale assessments to an independent, blinded reviewer

**Statistical methods:** This is a Phase I trial, with safety as the primary measure. Sample size was not determined through statistical justification.

# 3 TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES TABLE OF CONTENTS

| 1 | | ADMINISTRATIVE INFORMATION | 2 |
|----|------|--------------------------------------------------------|----|
| | 1.1 | Summary of Changes | 2 |
| | 1.2 | Contact Information | |
| 2 | | SYNOPSIS | |
| 3 | | TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES | 12 |
| | TABI | LE OF CONTENTS | |
| | LIST | OF TABLES | 15 |
| | LIST | OF FIGURES | 15 |
| 4 | | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 16 |
| 5 | | INTRODUCTION | 18 |
| | 5.1 | Background and Preliminary Data | 18 |
| | 5.2 | Rationale for Gene Transfer to SMA Type 1 Patients | 18 |
| | 5.3 | Non-Clinical Studies | 21 |
| 6 | | TRIAL OBJECTIVES AND PURPOSE | 24 |
| | 6.1 | Primary Objective | 24 |
| | 6.2 | Secondary Objectives. | 24 |
| | 6.3 | Exploratory Objectives | 24 |
| 7 | | INVESTIGATIONAL PLAN | 25 |
| | 7.1 | Overall Study Design | 25 |
| | 7.2 | Number of Subjects | 25 |
| | 7.3 | Treatment Assignment | 26 |
| | 7.4 | Criteria for Study Termination. | 26 |
| 8 | | SELECTION AND WITHDRAWAL OF SUBJECTS | 30 |
| | 8.1 | Subject Inclusion Criteria | 30 |
| | 8.2 | Subject Exclusion Criteria | 30 |
| | 8.3 | Subject Withdrawal Criteria | 31 |
| 9 | | TREATMENT OF SUBJECTS | 31 |
| | 9.1 | Description of Study Drug | 31 |
| | 9.2 | Concomitant Medications | 32 |
| | 9. | 2.1 Prophylactic Administration of Prednisolone | 32 |
| | 9. | 2.2 Prohibited Medications | 33 |
| 10 | | STUDY DRUG MATERIALS AND MANAGEMENT | 33 |
| | 10.1 | Study Drug | 33 |
| | 10.2 | Study Drug Packaging and Labeling | 33 |
| | 10.3 | Study Drug Storage | 33 |
| | 10.4 | Study Drug Preparation | 33 |

| 10.5 | Administration | | 35 |
|-------|----------------------|-----------------------------------|----|
| 10.6 | Dose Escalation | | 35 |
| 10.7 | Study Drug Accoun | ntability | 36 |
| 10.8 | Study Drug Handlin | ng and Disposal | 36 |
| 11 | ASSESSMENTS | | 36 |
| 11.1 | Safety Parameters | | 36 |
| 11. | .1 Dose Limitii | ng Toxicity | 36 |
| 11. | .2 Discontinuat | tion Rules | 37 |
| 11.2 | Demographic/Medic | cal History | 37 |
| 11.3 | Vital Signs | | 37 |
| 11.4 | Pulse Oximetry | | 37 |
| 11.5 | Weight and Height. | | 37 |
| 11.6 | Physical Examination | on | 37 |
| 11.7 | Vaccination Recomm | mendations | 38 |
| 11.8 | Physical Therapy As | ssessments | 38 |
| 11.8 | .1 CHOP-INTE | END | 38 |
| 11.8 | Bayley Scale | e of Infant Development version 3 | 38 |
| 11.9 | | stones Checklists | |
| 11.10 | Video Evidence | | 39 |
| 11.11 | ACTIVE-mini | | 39 |
| 11.12 | Electrophysiology A | Assessments | 39 |
| 11. | | | |
| 11. | 2.2 CMAP | | 40 |
| 11. | 2.3 MUNE | | 40 |
| 11.13 | Chest X-ray | | 40 |
| 11.14 | Swallowing Test | | 40 |
| 11.15 | Echocardiography | | 40 |
| 11.16 | Electrocardiogram ( | (ECG) | 40 |
| 11.17 | Pulmonary Assessm | nent | 40 |
| 11.18 | | usion Site | |
| 11.19 | | nents | |
| 11. | 9.1 Hematology | 7 | 42 |
| 11. | | nistry | |
| 11. | 9.3 Urinalysis | | 42 |
| 11. | | Studies | |
| 11. | | lood Gas | |
| 11. | | ogy | |
| 11. | | nmunology Blood | |

| | 11.19.8 | Baseline Screening of Mother | 43 |
|---|---|---|---|
| | 11.19.9 | IFN-γ ELISpots | 43 |
| | 11.19.10 | Research Blood Sample | 43 |
| | 11.19.11 | Saliva, Urine, and Stool Collection. | 43 |
| 12 | ADVE | RSE AND SERIOUS ADVERSE EVENTS | 44 |
| | 12.1 Def | inition of Adverse Events | 44 |
| | 12.1.1 | Adverse Event (AE) | 44 |
| | 12.1.2 | Serious Adverse Event (SAE) | 44 |
| | 12.1.3 | Other Adverse Event (OAE) | 44 |
| | 12.2 Rela | ationship to Study Drug | 44 |
| | 12.3 Rec | ording Adverse Events | 45 |
| | 12.4 Rep | orting Adverse Events | 45 |
| 13 | DATA | SAFETY MONITORING BOARD | 46 |
| | 13.1 DSN | MB Reporting and Meetings | 46 |
| | 13.2 DSN | MB Membership | 47 |
| 14 | STATIS | STICS | 47 |
| 15 | DIREC | T ACCESS TO SOURCE DATA/DOCUMENTS | 48 |
| | 15.1 Stud | dy Monitoring | 48 |
| | 15.2 Aud | lits and Inspections | 48 |
| | 15.3 Inst | itutional Review Board (IRB) | 48 |
| | 15.4 Qua | lity Control and Quality Assurance | 48 |
| 16 | ETHIC | S | 49 |
| | 16.1 Ethi | cs Review | 49 |
| | 16.2 Ethi | cal Conduct of the Study | 49 |
| | 16.3 Wri | tten Informed Consent | 49 |
| 17 | DATA | HANDLING AND RECORDKEEPING | 49 |
| | 17.1 Elec | etronic Case Report Forms | 49 |
| | 17.2 Insp | pection of Records | 50 |
| | 17.3 Rete | ention of Records. | 50 |
| | 17.4 Rete | ention of Samples | 50 |
| 18 | PUBLIC | CATION POLICY | 50 |
| 19 | LIST O | F REFERENCES | 52 |
| 20 | APPEN | DICES | 54 |
| | Appendix 1 | Declaration of Helsinki: Ethical Principles for Medical Research | . ـ |
| | | blving Human Subjects | |
| | Appendix 2 | Autopsy Plan | |
| | Appendix 3 | Chop-intend. | |
| | Appendix 4 | Bayley Scale of Infant Development version 3: Gross and Fine Mols Subparts and Speech and cognition subparts | otor<br>65 |

| e | | 1 |
|---|---|---|
| Appendix 5 | Gross Motor Skills Checklist | 81 |
| | LIST OF TABLES | |
| Table 1 | Summary of Protocol Section Changes and Additions | 2 |
| Table 2 | Important Study Contact Information | |
| Table 3: | Study Vendor Listing | |
| Table 4 | Abbreviations and Specialist Terms | |
| Table 5 | Spinal Muscular Atrophy Classification | |
| Table 6 | Schedule of Assessments | |
| Table 7 | Investigational Product | 32 |
| Table 8 | Total Dose | |
| Table 9 | Adverse Event Classification | 37 |
| Table 10 | Motor Milestone Development Survey | 38 |
| Table 11 | Total Blood Volume | 41 |
| Table 12 | Tissue Samples for Analysis | 60 |
| | LIST OF FIGURES | |
| Figure 1 | Kaplan-Meier survival curves and survival probabilities for SMA 7 2, and 3 | Гуре 1,<br>20 |
| Figure 2 | Study results, including staining of transduced spinal motor neuron expression levels, righting ability, and weight and survival curves. | |
| Figure 3 | Body mass of treated and control mice showed no difference | |
| Figure 4 | Study Design | 27 |

# 4 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

The following abbreviations and specialist terms are used in this study protocol.

Table 4 Abbreviations and Specialist Terms

| Abbreviation or Specialist Term | Definition |
|---|---|
| ACTIVE | Ability Captured Through Interactive Video Evaluation |
| AE | Adverse event |
| Alk Phos | Alkaline Phosphatase |
| ALT | Alanine Aminotransferase |
| AST | Aspartate Aminotransferase |
| BiPAP | Non-invasive Positive Pressure Ventilator |
| BUN | Blood urea nitrogen |
| CBER | Center for Biologics Evaluation and Research |
| CHOP-INTEND | Children's Hospital of Philadelphia Infant Test of Neuromuscular<br>Disorders |
| CK | Creatine kinase |
| CMAP | Compound Muscle Action Potentials |
| cmm | Cubic millimeter |
| DLT | Dose Limiting Toxicity |
| DRP | DNAse-Resistant Particle. Titer is based off the original certificate of analysis |
| DSMB | Data Safety Monitoring Board |
| ЕСНО | Echocardiogram |
| eCRF | Electronic Case Report Form |
| EIM | Electrical Impedance Myography |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| HIPAA | Health Insurance Portability and Accountability Act |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| ICJME | International Committee of Medical Journal Editors |
| IEC | Independent Ethics Committee |
| IND | Investigational New Drug |
| IRB | Institutional Review Board |
| mo | months |

| Abbreviation or Specialist Term | Definition |
|---|---|
| MUNE | Motor Unit Number Estimation |
| NHP | Non-human primate |
| OAE | Other significant adverse event |
| PI | Principal Investigator. The investigator who leads the study conduct at an individual study center. Every study center has a principal investigator. |
| SAE | Serious adverse event |
| scAAV | Self-complimentary adeno-associated virus |
| SMA | Spinal muscular atrophy |
| SMN | Survival motor neuron |
| WT | Wild type. Wild type mice are those not affected with SMA. |
| yo | Years old |

# 5 INTRODUCTION

This is the first clinical gene therapy trial for spinal muscular atrophy (SMA). The SMN gene will be transferred using self-complementary adeno-associated virus (scAAV) type 9 under control of the chicken-β-actin hybrid promoter. Pre-clinical studies have demonstrated survival of the SMN-Δ7 mouse model for SMA from a median of 15.5 days to over 1 year, following intravenous delivery to the facial vein. This clinical trial is an open-label, single injection ascending dose study in which AVXS-101 will be delivered one-time through a venous catheter inserted into a peripheral vein (arm, leg, or scalp) in SMA Type 1 subjects with 2 copies of SMN2.

# 5.1 Background and Preliminary Data

Spinal muscular atrophy is a neurogenetic disorder caused by a loss or mutation in the survival motor neuron 1 gene (SMN1) on chromosome 5q13, which leads to reduced SMN protein levels and a selective dysfunction of motor neurons. SMA is an autosomal recessive, early childhood disease with an incidence of 1:11,000 live births. 14 SMA is the leading cause of infant mortality due to genetic diseases. Disease severity and clinical prognosis depends on the number of copies of SMN2. In its most common and severe form (Type 1), hypotonia and progressive weakness are recognized in the first few months of life, leading to diagnosis by 6 months of age and then death due to respiratory failure by age two. SMA Type 1 is the leading genetic cause of infant death. Motor neuron loss in SMA Type 1 is profound in the early postnatal period (or may even start in the pre-natal period), whereas motor neurons in Type 2 and 3 SMA patients adapt and compensate during development and persist into adult life. The findings from various neurophysiological and animal studies have shown an early loss of motor neurons in the embryonic and early postnatal periods. <sup>10,11,12</sup> From a clinical perspective, these findings emphasize the importance of targeting the SMA Type 1 group for gene transfer of SMN2 in hopes of rescuing neurons at this critical stage. Our goal is to modify the SMA Type 1 phenotype, which will hopefully lead to a milder disease course and prolonged survival as seen in SMA Type 2 and 3 patients.

Therapeutic efforts in SMA have focused on the potential for small molecules to increase SMN levels. These include deacetylase inhibitors, such as, valproic acid, sodium butyrate, phenylbutyrate, and trichostatin A. These agents activate the SMN2 promoter, resulting in increased full-length SMN protein in SMA animal models. However, clinical trials employing several of these agents, most notably phenylbutyrate, valporic acid, and hydroxyurea, have not resulted in clinical benefit (www.ClinicalTrials.gov, and Darbar, et al<sup>17</sup>). A dose escalation trial of scAAV9.CB.SMN will provide information for the potential gene transfer has in treating Type 1 SMA patients and will hopefully show promise for success in modifying the disease prognosis. This will be a dose escalation study that includes 15 Type 1 patients with 2 copies of SMN2.

# 5.2 Rationale for Gene Transfer to SMA Type 1 Patients

We have chosen Spinal Muscular Atrophy (SMA) Type 1 as the target for this gene therapy study. We believe there is a strong rationale for this based on studies of the natural history of this disease. The classification of SMA is shown below (Table 5); Type 0 to Type 4 SMA is described. SMA is conventionally classified into four phenotypes on the basis of age of onset

and highest motor function achieved, with an additional phenotype (type 0) to describe the severe forms of antenatal-onset spinal muscular atrophy.<sup>1,2</sup>

 Table 5
 Spinal Muscular Atrophy Classification

| Туре | Age at Onset | Highest Function | Natural Age at Death | SMN2 No. |
|---|---|---|---|---|
| 0 | Prenata <b>l</b> | Respiratory support | <1 mo | 1 |
| 1 | 0 <b>-</b> 6 mo | Never sit | <2 y | 2 |
| 2 | <18 mo | Never stand | >2 y | 3, 4 |
| 3 | >18 mo | Stand alone | Adult | |
| 3a | 18 mo-3 y | Stand alone | Adult | 3, 4 |
| 3b | >3 v | Stand alone | Adu <b>l</b> t | 4 |
| 4 | >21 v | Stand alone | Adu <b>l</b> t | 4-8 |

SMA Type 1 patients by definition never attain independent sitting and have hypotonia within the first 6 months of life. SMA Type 1 is the leading genetic cause of infant death. In contrast, SMA Type 2 manifests within the first 18 months, and children afflicted with this condition are able to maintain sitting unassisted but never walk independently. SMA Type 3 patients attain the ability to walk unaided [Type 3a have onset <3yo; Type 3b have onset >3 yo]. SMA Type 4 is an adult onset disease. The genetic cause for SMA is well established and is intimately involved with one's prognosis. All forms of SMA are autosomal recessive in inheritance and are caused by mutations of the survival motor neuron 1 (SMN1) gene. Humans also carry a second nearly identical copy of the SMN1 gene called SMN2.<sup>3</sup> Both the SMN1 and SMN2 genes express SMN protein, however, the amount of functional full-length protein produced by SMN2 is much less (by 10-15%) than that produced by SMN1.<sup>3-5</sup> Although SMN2 cannot completely compensate for the loss of the SMN1 gene, patients with milder forms of SMA generally have higher SMN2 copy numbers. 6-7 Quantitative analysis of SMN2 copies in 375 patients with Type 1, Type 2, or Type 3 SMA showed a significant correlation between SMN2 copy number and SMA type, as well as, duration of survival. 80% of patients with Type 1 SMA carry one or two SMN2 copies, 82% of patients with Type 2 SMA carry three SMN2 copies, and 96% of patients with Type 3 SMA carry three or four SMN2 copies.<sup>8</sup> Among 113 patients with Type 1 SMA, 9 with one SMN2 copy lived <11 months, 88/94 with two SMN2 copies lived <21 months, and 8/10 with three SMN2 copies lived 33–66 months. Even more refined data, describing this relationship, has been generated and has also influenced our choice of the study target group. The median survival for patients with SMA Type 1 is 7.4 months with the age of onset being the most predictive factor in survival.9

The severity of SMA type 1 is unequivocally demonstrated by prognosis as illustrated in Kaplan-Meier survival curves shown in Figure 1.

Figure 1 Kaplan-Meier survival curves and survival probabilities for SMA Type 1, 2, and 3



In Figure 1, the relative stability of the clinical course of SMA Types 2 and 3 is dramatically illustrated. Perhaps most importantly these findings show that outcome differences are related to the number of SMN2 copies that enable motor neurons to adapt and compensate during the growth of the child and persist into adult life. This contrasts with SMA Type 1 where motor neuron loss is profound in the early postnatal period (or may even start in the pre-natal period, especially for SMA Type 1 patients presenting in first three months of life). The findings in Figure 1 confirm other pieces of evidence from neurophysiological studies and animal studies that also show early loss of motor neurons in the embryonic and early postnatal periods. <sup>10,11,12</sup> From a clinical trials perspective these findings emphasize the importance of targeting SMA Type 1 for gene transfer of SMN2 in hopes of rescuing neurons at this critical stage. Ultimately, the goal is to modify the SMA Type 1 phenotype leading to a milder course and prolonged survival, as we see in SMA Type 2 or 3 patients.

These findings more clearly provide the rationale for a clinical gene transfer trial in the younger patients making it more difficult to justify even Phase I safety trials in older (SMA Type 2 or 3) subjects. Based upon what we know about the natural history of SMA, gene transfer in the older, less severe SMA types (2, 3, and 4), is less likely to have a significant, clinical effect than it would in the younger Type 1 patients. Since the motor neuron pool is stable in older patients due to higher copy number of SMN2, asking Type 2, 3, or 4 patients to undergo safety trials with possibly only minimal benefit is highly unreasonable. It is much more appropriate and safe to prove tolerability in the younger SMA Type 1 group, in which death is the unequivocal outcome. Also, the poor prognosis of the SMA Type 1 patients, who only have 2 copies of SMN2, warrants the rescue of their lives as our top priority at this time.

Factors other than risk-benefit discourage Phase I trials in older SMA patients. The gene transfer viral dose for older patients, which is based on body weight, is much greater than what would be needed for an infant. Not only does this add significantly to the cost of the clinical trial, in some

cases, it could exceed the capacity of the vector manufacturing facility. These added costs, in addition to an increased risk prior to an established proof of principle provide a clear rationale for treating the younger Type 1 patients who have only 2 copies of SMN2. Also present is the issue of a greater chance of encountering pre-existing immunity to AAV in these older, Type 2 and 3 patients.

We also have good reason to believe that there are very few safety issues to be concerned about when targeting the SMA Type 1 group for this clinical gene therapy trial. Overexpression of SMN has been shown to be well tolerated in both mice and non-human primates, and in humans high copy number of SMN2 poses no risk (as seen in Type 2, 3, and 4 patients who have high SMN2 copy number). This allows us to utilize robust, ubiquitous expression systems (like the CB-promoter) to ensure sustained, high-level SMN expression. Additionally, it is important to point out that recombinant scAAV can be employed for this trial because of the small size of the SMN gene. This enables efficient packaging and allows for efficient gene transfer with lower viral titers (a safety consideration), compared with prototypical single-stranded AAV vectors.

Our recent studies using scAAV9.CB.SMN show a robust postnatal rescue of SMA mice with correction of motor function, neuromuscular electrophysiology and survival after a onetime delivery of vector. <sup>13</sup> Intravenous scAAV9 is able to transduce neurons, muscle and vascular endothelium, all of which have been proposed as target cells for SMA treatment.

Taken altogether, our preclinical efficacy and toxicology studies in mice and non-human primates have increased our confidence that our Phase Ib trial will be safe and will have a high potential for success in treating this devastating disease.

# **5.3** Non-Clinical Studies

A mouse model was developed by the Arthur Burghes Laboratory after a generation of multiple variants. It was found that the double transgenic, referred to as the SMN- $\Delta$ 7 mouse, provided the most suitable model to study gene transfer. 18 Studies performed in the Kaspar laboratory have shown that injecting 5 X 10<sup>11</sup> viral genomes of scAAV9.CB.SMN into the facial vein on day 1 old mice rescues the SMN-Δ7 mouse model. <sup>13</sup> Figure 2 shows the results of these studies, including staining of transduced spinal motor neurons, SMN expression levels, righting ability, and weight and survival curves. Approximately  $42 \pm 2\%$  of lumbar spinal motor neurons were transduced in scAAV9.CB.SMN treated mice. SMN levels were increased as well, in brain, spinal cord, and muscle of scAAV9.CB.SMN-treated animals, compared to untreated SMA mice (although lower than WT controls). SMA animals treated with either scAAV9.CB.SMN or scAAV9.CB.GFP on P1 were assessed for their righting ability and were compared to WT control mice and untreated mice. WT controls could right themselves quickly, whereas the SMN- and GFP-treated SMA animals showed difficulty at P5. However, by P13, 90% of SMNtreated animals could right themselves compared with 20% of GFP-treated controls and 0% of untreated SMA animals. At P18, SMN-treated animals were larger than GFP-treated animals, but smaller than WT controls. Locomotive ability of the SMN-treated mice was nearly identical to WT controls, as assayed by open field testing and wheel running.

Survival of SMN-treated SMA animals compared with GFP-treated SMA animals was significantly improved. No GFP-treated control animals survived past P22 and had a median life span of 15.5 days. The weights of GFP mice peaked at P10 and then precipitously declined until death, while SMN mice showed a steady weight gain until around P40 with it stabilizing at 17g

(about half the weight of WT controls). The smaller size of corrected animals is likely related to the tropism and incomplete transduction of scAAV9, resulting in a 'chimeric' animal in which some cells were not transduced. Additionally, the smaller size suggests an embryonic role for SMN. Most remarkably, SMN-treated mice survived well past 250 days of age.

Figure 2 Study results, including staining of transduced spinal motor neurons, SMN expression levels, righting ability, and weight and survival curves



- a) Shows transduced motor neurons in lumbar spinal cord
- b) Western Blots of SMN expression in CNS and muscle
- Improved righting ability of SMN-treated- similar to WT controls by P13
- d) SMN- treated are larger than GFP-treated at P18
- e) Survival of SMN-treated markedly improved compared to GFP- treated
- f) Body weight increased in SMNtreated vs GFP

Toxicology biodistribution studies were generated by the Kaspar laboratory. In the non-GLP studies, 24 mice and 4 non-human primates (NHPs) were injected, by way of vascular delivery, with scAAV9.CB.SMN. To assess toxicity and safety scAAV9.CB.SMN was injected into P1 wild type FVB mice with either vehicle (PBS) (3 males/6 females) or  $3.3 \times 10^{14} \text{ vg/kg}$  of scAAV9.CB.SMN (6 males/9 females) via the facial temporal vein. This dose was previously shown to be most efficacious in the  $\Delta 7$  mouse model of SMA16. P1 mice were used in anticipation of simulating potential clinical studies in infants, which is the planned population for the first-in-human clinical trial. All mice survived the injection procedure and the initial 24-hour observation period without any signs of distress or weight loss. Body mass was measured and hands-on observations were performed weekly for the remainder of the study; neither revealed any difference between control and treated cohorts (Figure 3).

Figure 3 Body mass of treated and control mice showed no difference



At 60, 90 and 180 days post-injection, blood from the mice was collected for hematology studies and clinical chemistries assessment (ALT, AST, ALK Phos, creatinine, BUN, electrolytes, and CK). All were normal except for one variant at the 90 day time point. This difference appeared to be due to a technical problem relating to the site of blood draw, which differed from that of all other mice. For histopathology, 13 mice were necropsied at 120 days post-injection and 8 mice at 180 days. All organs were normal; in particular there was no inflammation seen in any section from any organ (heart, liver, kidney, muscle, gonads, brain, lung, lymph nodes, and intestines).

In the safety study for the four male Cynomolgus Macaques, subjects were injected at 90 days of age to closely mimic the likely age of administration of treatment in SMA Type 1 infants. The scAAV9.CB.SMN vector was administered one time by catheterization of the saphenous vein with a dose of 6.7 x 10<sup>13</sup>/kg, which corresponds to the lowest dose tested for which SMN-Δ7 mice showed a significant increase of survival. Animals were followed for six months until they were sacrificed at approximately 9 months of age. No adverse effects were seen, and all clinical chemistries were normal. T-cell immune response was tested using ELISpot in peripheral blood mononuclear cells (PBMCs), and all were negative at 6 months post injection.

These mouse and monkey studies can be summarized as follows. The serum chemistry and hematology studies were unremarkable as was the histopathology assessment. The NHP subjects mounted appropriate immune responses to capsid (but not to transgene), with very high transgene expression persisting at 6 months post-injection. In conclusion, these studies provide strong evidence that systemically-delivered scAAV9.CB.SMN is safe and well tolerated, even at the high doses required for penetration of the blood-brain barrier.<sup>13</sup>

Formal IND-enabling GLP pharmacology, toxicology, and biodistribution studies were discussed with the FDA at the Pre-IND meeting held January 2012. The toxicology plan discussed with CBER was found to be acceptable for the initiation of this Phase I trial.

# 6 TRIAL OBJECTIVES AND PURPOSE

# 6.1 Primary Objective

The primary outcome for this clinical trial is safety. Discontinuation criteria are based on the development of unacceptable toxicity, defined as the occurrence of any one Grade III or higher, unanticipated, treatment-related toxicity that presents with clinical symptoms and requires medical treatment.

# 6.2 Secondary Objectives

A secondary outcome will include time from birth to either (a) requirement of  $\geq$ 16-hour respiratory assistance per day (includes BiPAP) continuously for  $\geq$ 2 weeks in the absence of an acute reversible illness, excluding perioperative ventilation or (b) death.

Secondary outcomes will also include the change in CHOP-INTEND from baseline score and demonstration of improvement of motor function and muscle strength as determined by achievement of significant development milestones including but not limited to the ability to sit alone and roll over unassisted. Additionally, sponsor may choose to provide videos of the physical exams, CHOP-INTEND assessments, and/or Bayley Scale assessments to an independent, blinded reviewer for confirmation of the development milestones.

# 6.3 Exploratory Objectives

Exploratory outcome measures will be tested during the study as part of the program and product development plan; however if exploratory measurement results show efficacy and primary outcomes do not reach statistical significance, the only interpretation is that the results show a trend toward benefit but can never supersede primary measures. These exploratory outcome measures will include:

- ACTIVE-mini (Ability Captured Through Interactive Video Evaluation-mini) evaluation of infant movement ability.
- Patient functional measures using the Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP-INTEND). This test has been studied and validated in infants with spinal muscular atrophy and was found to be reliable in this population.<sup>19</sup>
- Bayley Scale of Infant Development version 3 is a standardized, norm-referenced infant assessment. The gross and fine motor portions as well as speech and cognition portions of this test will administered if the child reaches or exceeds a score of 60 out of 64 on the CHOP-INTEND.
- Motor neuron function will be assessed via evoked compound motor action potentials (CMAP) and motor unit number estimation (MUNE).
- Pathological status of muscles will be quantified by Electrical Impedance Myography (EIM).
- The age at which significant motor milestones are achieved will be assessed using a standard Motor Milestone Development Survey shown in Table 10 in Section 11.1.10.
- Compelling, demonstrable, documented evidence of efficacy as determined by changes in functional abilities as captured during videotaping sessions during site visits and/or captured by subject/parent/legal guardian at home.

# 7 INVESTIGATIONAL PLAN

# 7.1 Overall Study Design

The proposed clinical trial is an open-label, single injection ascending dose study of self-complementary AAV9 carrying the SMN gene under the control of a hybrid CMV enhancer/chicken AVXS-101 delivered one-time through a venous catheter inserted into a peripheral vein (arm, leg, or scalp) of Type 1 spinal muscular atrophy subjects.

The primary analysis for efficacy will be assessed when all patients reach 13.6 months of age (a database lock will be performed at the time point at which all patients reach 13.6 months of age). A follow-up safety analysis will be completed at the time point at which the last patient reaches 24 months post-dose.

This dose escalation study involves four cohorts. There will be at least a 3 week intra-cohort dosing interval between dosing of patients within a cohort to allow review of the safety analysis from five time points (days 1, 2, 7, 14, and 21) prior to dosing of the next patient. There will be at least a 4-week inter-cohort dosing interval between dosing of patients between cohorts to allow time for review of the safety analysis of at least six time points (days 1, 2, 7, 14, 21, and 30) from all the patients within a cohort. Safety analysis will be done by the investigators and the DSMB, as well as, time for decisions to be made about whether to implement a higher dose group. Dose escalation will be based on dose-limiting toxicity (DLT).

Cohort 1 will consist of three (3) SMA patients followed by Cohort 2A with a minimum of three (3) and no more than six (6) SMA patients to receive a single infusion at escalating doses.

- Cohort 1 (Low Dose): 6.7 X 10<sup>13</sup> vg/kg (n=3)
- Cohort 2A (Intermediate Dose):  $2.0 \times 10^{14} \text{ vg/kg}$  (n $\geq 3$  and n $\leq 6$ )

Cohort 2B and Cohort 3 will each consist of three (3) SMA patients to receive a single infusion at escalating doses.

- Cohort 2B: 2.0 X 10<sup>14</sup> vg/kg (n=3)
- Cohort 3 (High Dose): 3.3 X 10<sup>14</sup> vg/kg (n=3)

Cohort 2B will be done first and if efficacy is favorable but does not fully improve subjects to normal, Cohort 3 at high dose will be implemented.

Treatment of Cohort 3 is permitted based on safety assessment presented in the IND. A score of 8 or higher on the Bayley Scales of Infant Development will be considered the low end of normal. If efficacy (defined as any clinical improvement from baseline of either primary or exploratory outcome measures) is observed at the intermediate dose (2.0 X 10<sup>14</sup> vg/kg), the Principal Investigator may continue to enroll at the intermediate dose up to a maximum of 9 patients.

If no clinically significant improvement without toxicity is observed, the possibility of adding an additional escalation cohort at a higher dose will be discussed with the FDA, DSMB and relevant oversight regulatory agencies.

# 7.2 Number of Subjects

A total of 15 subjects may be enrolled.

# 7.3 Treatment Assignment

This is an open-label study. Treatment will be assigned in accord with the dose escalation schedule specified in Section 10.6.

# 7.4 Criteria for Study Termination

An independent Data Safety Monitoring Board (DSMB) and safety monitor will monitor safety data on a continual basis throughout the trial. The DSMB can recommend early termination of the trial for reasons of safety. Study enrollment will be halted by the investigators when any subject experiences a Grade III, or higher adverse event toxicity that is unanticipated and possibly, probably, or definitely related to the study drug that presents with clinical symptoms and requires medical treatment. This will include any patient death, important clinical laboratory finding, or any severe local complication in the injected area related to administration of the study agent. If after review by the DSMB, IRB, IBCSC, NIH-OBA and FDA, the decision is made to continue, the study will proceed according to the dose escalation schedule.

Subjects may be discontinued from further study participation or the trial may be terminated for the following reasons:

- Development of unacceptable toxicity, defined as the occurrence of any one Grade III or higher, unanticipated, treatment-related toxicity that presents with clinical symptoms and requires medical treatment.
- Patient requires at least 16-hour per day of ventilation support for breathing, including BiPAP use, for ≥14 consecutive days in the absence of an acute reversible illness, excluding perioperative use
- Death
- Failure to comply with protocol-required visits or procedures
- Study is terminated by sponsor
- Subject withdrawal of consent to participate further

AveXis, Inc.

Investigational Product: AVXS-101

Protocol Number: AVXS-101-CL-101 Protocol Version 14.0 / 21 Apr 2016



 Table 6
 Schedule of Assessments

| | Baseline | Vector Infusion | | | | Follow Up Year 1 | | | | | | | Follow Up Year 2 | | | Long Term<br>Monitor | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Interval | Screening | (Inpatient) | | | (Outpatient) | | | | | | | | | | | | | |
| Visit | 1 | | 2 | | | 3 | 4 | 5 | 6 | 7 | 8 | Monthly | Every 3<br>Months | Every 6<br>Months | Every<br>Month <sup>g</sup> | Every Q3 Q6<br>Month <sup>9</sup> Months Months | | Annually |
| Days in Study <sup>a</sup> | -30 (± 7) | -1 | 0 | 1 | 2 | 7 | 14 | 21 | 30 | 60 | 90 | Up to 12 Months | | 13-24 Months | | Through<br>15 years | | |
| Informed Consent | х | | | | | | | | | | | | | | | | | |
| Chest X-Ray | х | | | | | | | | | | | | | | | | | |
| Medical History | х | | | | | | | | | | | | | | | | | |
| Physical Exam +<br>Vitals | х | Χc | Χď | х | х | х | х | х | х | х | х | х | х | х | Χa | х | х | х |
| Pulmonary<br>Assessment | х | | | х | | х | х | х | х | х | х | х | х | х | Χa | х | х | х |
| Photograph<br>Injection site | х | х | х | x | х | х | х | х | х | х | х | х | х | x | Χa | х | х | |
| Swallowing Test | х | | | | | | | | | | | | | х | | | х | |
| Pulse Oximetry <sup>d</sup> | х | х | х | х | х | х | Х | х | х | Х | х | х | х | х | Χg | х | х | |
| Capillary Blood Gas | х | х | х | х | х | | | | | | | | | | | | | |
| Safety Labs (Blood) | х | х | | х | х | х | Х | х | Х | Х | х | | х | х | Χg | х | Х | |
| Coagulation Studies (PT/INR/PTT) | | | | | | | | | | | х | | х | х | | х | х | |
| Safety Labs<br>(Urinalysis) | х | х | | х | х | х | х | | х | | х | | х | х | Χg | х | х | |
| Immunology<br>(AntiAAV9/SMN Ab<br>& T-Cells) | x | | | | | х | х | х | х | х | х | | х | х | | х | x | |
| Research Blood <sup>e</sup> | х | | | | | | | х | х | х | х | | х | х | | х | Х | |
| CHOP-INTEND <sup>f</sup><br>(with video) | х | х | | | | | | | х | х | х | х | х | х | Xa | х | х | |

| Study Interval | Baseline | Ved | ctor Ir | nfusi | on | | Follow Up Year 1 | | | | | | | Fallow Un Vaca 2 | | | Long Term | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Interval | Screening<br>1 | (Inpatient) | | | (Outpatient) | | | | | | | | Follow Up Year 2 | | | Monitor | | |
| Visit | | | | | 3 | 4 | 4 5 | 6 | 7 | 8 | Monthly | Every 3<br>Months | Every 6<br>Months | Every<br>Month <sup>g</sup> | Q3<br>Months | Q6<br>Months | Annually | |
| Days in Study <sup>a</sup> | -30 (± 7) | -1 | 0 | 1 | 2 | 7 | 14 | 21 | 30 | 60 | 90 | U | Up to 12 Months 13-24 Months | | 13-24 Months | | Through<br>15 years | |
| Bayley <sup>b</sup> | х | х | | | | | | | х | х | х | Xp | Хp | Χp | Χg | х | х | |
| ACTIVE-mini | х | Х | | | | х | х | х | Х | х | х | х | х | х | | х | х | |
| CMAP/MUNE/EIM | х | | | | | | | | Х | | х | | х | х | | х | х | |
| Research Urine | х | | | х | х | х | Х | х | Х | Х | х | х | х | х | | х | х | |
| Research Saliva & Stool | х | | | х | х | х | х | х | х | х | х | х | х | х | | х | х | |
| Development<br>Milestones/Gross<br>Motor Skills<br>Checklist (with<br>video) | х | | | | | | | | x | | | | | x | Xa | х | | х |
| ECHO/ECG | х | | | | | | | | Х | | | | | х | | х | | Х |
| Prednisolone<br>Dosing | | Х | x | х | х | х | х | | | | | | | | | | | |
| Gene Transfer | | | х | | | | | | | | | | | | | | | |
| Adverse Events | Х | х | Х | Х | Х | Х | х | Х | х | Х | х | х | Х | х | Χg | Х | Х | Х |
| Concomitant<br>Medications | | To be collected from 2 weeks before study dose until final study visit, recorded on separate CRF | | | | | | | | | | | х | | | | | |

a Visits on Days 7, 14 and 21 allow a window of ±2 days; all monthly visits following (Visit 6 to 29) allow a window of ±7 days.

b The gross and fine motor portions of this test will be administered monthly through 14 months post-dose if a patient reaches or exceeds a score of 60 out of 64 on the CHOP-INTEND. The cognition portion of this test will be administered every three months if a patient reaches or exceeds a score of 60 out of 64 on the CHOP-INTEND. CHOP-INTEND assessment will be discontinued and only the Bayley will be administered for subjects that achieve two consecutive scores of 64.

c Vital signs recorded every four (4) hours during inpatient hospitalization.

d Continuous monitoring during gene transfer procedure. Axillary temperature to be captured pre- and post- infusion.

e Research blood sample will be used to perform baseline exon 7 modification testing and could also be used to re-confirm SMA Type 1 diagnosis, SMN2 copy number, and exon-7 modification testing through a third-party laboratory.

f Subjects that achieve two consecutive scores of ≥62 may cease further CHOP-INTEND assessments, as per PI, physical therapist, and sponsor decision.

g Subjects for whom the decision is made to continue CHOP-INTEND assessments, or who don't reach score ≥62, will continue to complete monthly visits during Year 2.

## 8 SELECTION AND WITHDRAWAL OF SUBJECTS

SMA Type 1 subjects, six months and younger with proven mutations of the SMN1 gene will be enrolled in this clinical trial. Patients will be of any racial, ethnic, or gender background. Enrollment will be staggered with at least 4 weeks between patient infusions. The assessment and full treatment plan will be used for all subjects in Cohort 2B (n=3) and potentially for subjects in Cohort 3 (n=6) to be included if subjects in Cohort 2B do not achieve a status of normal: a score of 8 or higher on the Bayley Scales of Infant Development will be considered the low end of normal.

# 8.1 Subject Inclusion Criteria

Subjects must meet all of the following Inclusion Criteria:

- 1. Six months of age and younger<sup>1</sup> at day of vector infusion with Type 1 SMA as defined by the following features:
  - a. Bi-allelic SMN1 gene mutations (deletion or point mutation) with two copies of SMN2 (no more and no fewer).
  - b. Patients 6 months and younger with a disease onset up to 6 months of age.
  - c. Hypotonia by clinical evaluation with delay in motor skills, poor head control, round shoulder posture and hypermobility of joints.
- First nine subjects enrolled under previous version(s) of the protocol could be nine months of age or younger. Inclusion revised to reflect six months of age or younger in 24 Jun 2015 Protocol Addendum #2.

Initial genetic testing and diagnosis completed at an institution/laboratory other than Nationwide Children's Hospital/Ohio State University is acceptable if proper documentation is received at Nationwide Children's Hospital, verified by the PI, and filed in the patient's medical record.

AveXis, Inc. may opt to confirm all genetic diagnoses through a contracted third-party laboratory utilizing an additional blood sample collected during a post-dose visit.

## 8.2 Subject Exclusion Criteria

Subjects must not meet any of the following Exclusion Criteria:

- 1. Active viral infection (includes HIV or serology positive for hepatitis B or C).
- 2. Use of invasive ventilatory support (tracheotomy with positive pressure)\* or pulse oximetry <95% saturation at the screening visit.
  - a. Patients may be managed using non-invasive ventilator support (BiPAP) for less than 16 hours a day at the discretion of their physician or research staff.
- 3. Concomitant illness that in the opinion of the PI creates unnecessary risks for gene transfer.
- 4. Concomitant use of any of the following drugs: drugs for treatment of myopathy or neuropathy, agents used to treat diabetes mellitus, or ongoing immunosuppressive therapy or immunosuppressive therapy within 3 months of starting the trial (eg, corticosteroids, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, intravenous immunoglobulin, rituximab).

5. Patients with Anti-AAV9 antibody titers >1:50 as determined by ELISA binding immunoassay.

- 6. Abnormal laboratory values considered clinically significant (GGT >3XULN, bilirubin ≥3.0 mg/dL, creatinine ≥1.8 mg/dL, Hgb <8 or >18 g/Dl; WBC >20,000 per cmm).
- 7. Participation in a recent SMA treatment clinical trial that in the opinion of the PI creates unnecessary risks for gene transfer.
- 8. Family does not want to disclose patient's study participation with primary care physician and other medical providers.
- 9. Patient with signs of aspiration based on a swallowing test and unwilling to use an alternative method to oral feeding.
- 10. Patients with c.859G>c modification in exon 7, based on predicted mild phenotype.

# 8.3 Subject Withdrawal Criteria

Subjects meeting the following criteria will be withdrawn:

- Development of unacceptable toxicity, defined as the occurrence of any one Grade III or higher, unanticipated, treatment-related toxicity that presents with clinical symptoms and requires medical treatment during the 2-year post-dose period
- Patient requires at least 16-hour per day of ventilation support for breathing, including BiPAP use, for 14 consecutive days in the absence of an acute reversible illness excluding perioperative use
- Death
  - Autopsies will be requested of any subjects that expire following participation in a gene transfer study as per the National Institutes of Health's Guidelines for Research Involving Recombinant or Synthetic Nucleic Acid Molecules; see Autopsy Plan in Appendix 2.
- Withdrawal of consent from further participation

Further guidance regarding determination of withdrawal criteria is outlined in Section 11.1.

## 9 TREATMENT OF SUBJECTS

Subjects will receive the gene transfer intravenous infusion under sterile conditions in a PICU patient room. The vector is formulated in the Nationwide Children's Investigational Pharmacy in approximately 10–20 mL/kg of normal saline and delivered to the PICU patient room in prelabeled syringes sealed in double leak-proof bags, carried in a designated lockable cooler.

The final formulated vector will be administered approximately at 10–20 mL/kg and slowly infused for approximately 60 minutes. The vector will be administered to the patient within 8 hours of preparation.

## 9.1 Description of Study Drug

The biological product is a non-replicating recombinant self-complementary adeno-associated virus serotype 9 (AAV9) containing the cDNA of the human SMN gene under the control of the cytomegalovirus (CMV) enhancer/chicken-β-actin-hybrid promoter (CB). The AAV inverted

terminal repeat (ITR) has been modified to promote intramolecular annealing of the transgene, thus forming a double-stranded transgene ready for transcription. This modified ITR, termed a "self-complementary" (sc) ITR, has been shown to significantly increase the speed of which the transgene is transcribed and the resulting protein is produced. The biological product, called scAAV9.CB.hSMN, expresses the human SMN protein.

Table 7 Investigational Product

| | Investigational Product |
|---|---|
| Product Name: | AVXS-101 |
| Dosage Form: 1.96 X 10 <sup>13</sup> DRP/mL (based off supercoiled qPCR) in either a 2 mL vial (with fill) or 5 mL vial (with 5 mL fill) All vials are screwcap polypropylene vials | |
| <b>(nit Dose</b> 10–20 mL/kg, in accord with dose escalation schedule | |
| Route of Administration | Peripheral vein intravenous infusion |
| Physical Description | AVXS-101 is provided in frozen 1 mL and 5 mL vials. Once thawed AVXS-101 is a clear liquid. |
| Manufacturer | Nationwide Children's Hospital Clinical Manufacturing Facility Center for Gene Therapy 700 Children's Drive Columbus, OH 43205 |

## 9.2 Concomitant Medications

Prior and concomitant medications will be captured in the eCRF from two weeks prior to study dosing through the last study visit.

# 9.2.1 Prophylactic Administration of Prednisolone

In every gene therapy study NCH has completed, including the first SMA patient, an antigen specific T-cell response to the AAV vector has been observed. This is an expected response between 2–4 weeks following gene transfer. One possible consequence to such antigen specific T-cell response is clearance of the transduced cells and loss of transgene expression. In an attempt to dampen the host immune response to the AAV based therapy, patients will be started on prophylactic prednisolone (glucocorticoid) (approximately 1 mg/kg/day) 24 hours prior to the gene transfer as agreed upon with FDA in the revised protocol submitted an IND update Serial No. 004, 31 Oct 2014. Treatment will continue for approximately 30 days with the following guidelines for tapering: When AST and ALT exceed 120 IU/L prednisolone will be maintained until enzymes fall below this level while at the same time monitoring T-cell response for decreases below 100 SFC per 10<sup>6</sup> PBMCs. Discrepancies from these precise recommendations will be at the discretion of the investigator based on potential safety issues for participating patients.

## 9.2.2 Prohibited Medications

Concomitant use of any of the use of any of the following medications is prohibited:

- Drugs for treatment of myopathy or neuropathy
- Agents used to treat diabetes mellitus
- Ongoing immunosuppressive therapy or immunosuppressive therapy within 3 months of starting the trial (e.g, corticosteroids, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, intravenous immunoglobulin, rituximab).

# 10 STUDY DRUG MATERIALS AND MANAGEMENT

AVXS-101 is manufactured in the cGMP facility of the Center for Gene Therapy at the Research Institute at Nationwide Children's Hospital. Only the number of vials required for stability testing and clinical retains will be stored at the cGMP facility.

# 10.1 Study Drug

AVXS-101

# 10.2 Study Drug Packaging and Labeling

Each vial is labeled with a specific log number and reagent code.

## 10.3 Study Drug Storage

AVXS-101 will be maintained at the Investigational Drug Service Pharmacy in the Hazardous Ultralow -80°C freezer located in room D01616 at NCH for the duration of the study.

# 10.4 Study Drug Preparation

Preparation of the gene vector will be done by the NCH research pharmacist according to the Manual of Operation Procedures. Immediately prior to transportation to the clinical setting, appropriate dilutions of the test article will be completed by the pharmacy. Documentation of the dilution will be completed by the pharmacy following standard pharmacy protocol. The vector will be diluted and manipulated in polypropylene syringes.

The vector is to be filled by the cGMP staff in screw cap vials at volumes of 5.0 mL (5 mL cryovial size) and 1.0 mL (2 mL cryovial size). The appropriate number of vials and volume of each will be determined for each patient based on body weight and specified dose cohort as illustrated in Table 8. The total vector genome dose will be calculated based on patient's body weight and rounded down to the closest 1 kg.

Protocol Number: AVXS-101-CL-101 Protocol Version 14.0 / 21 Apr 2016

AveXis, Inc. Investigational Product: AVXS-101

**Table 8** Total Dose

| Low Dose (6.7e13) vg/kg | | | | | | |
|---|---|---|---|---|---|---|
| Total Dose<br>(vg) | Vector Volume<br>(mL) | Total Volume (mL) | Syringe # | Syringe<br>Volume (mL) | Vector<br>Volume (mL) | Saline<br>Volume (mL) |
| 2.68E+14 | 13.7 | 67.3 | 1 | 33.7 | 6.8 | 26.8 |
| 2.00E+14 | 13.7 | 07.3 | 2 | 33.7 | 6.8 | 26.8 |
| 3.35E+14 | 17.1 | 84.2 | 1 | 42.1 | 8.5 | 33.5 |
| 3.33E±14 | 17.1 | 84.2 | 2 | 42.1 | 8.5 | 33.5 |
| 4.02E+14 | 20.5 | 101.0 | 1 | 50.5 | 10.3 | 40.3 |
| 4.02E+14 | 20.3 | 101.0 | 2 | 50.5 | 10.3 | 40.3 |
| 4.69E+14 | 22.0 | 117.9 | 1 | 58.9 | 12.0 | 47.0 |
| 4.09E+14 | 23.9 | 117.9 | 2 | 58.9 | 12.0 | 47.0 |
| | | | 1 | 44.9 | 9.1 | 35.8 |
| 5.36E+14 | 27.3 | 134.7 | 2 | 44.9 | 9.1 | 35.8 |
| | | | 3 | 44.9 | 9.1 | 35.8 |
| | | | 1 | 50.5 | 10.3 | 40.3 |
| 6.03E+14 | 30.8 | 151.5 | 2 | 50.5 | 10.3 | 40.3 |
| | | | 3 | 50.5 | 10.3 | 40.3 |
| | | | 1 | 56.1 | 11.4 | 44.7 |
| 6.7E+14 | 34.2 | 168.4 | 2 | 56.1 | 11.4 | 44.7 |
| | | | 3 | 56.1 | 11.4 | 44.7 |

| Intermediate Dose (2.0e14 vg/kg) | | | | | | | |
|---|---|---|---|---|---|---|---|
| Weight (kg) | Total Dose<br>(vg) | Vector Volume<br>(mL) | Total Volume<br>(mL) | Syringe # | Syringe Volume (mL) | Vector Volume<br>(mL) | Saline Volume<br>(mL) |
| 4 | 0.00E±14 | 40.9 | 67.2 | 1 | 33.7 | 20.4 | 13.3 |
| 4 | 8.00E+14 | 40.8 | 67.3 | 2 | 33.6 | 20.4 | 13.2 |
| 5 | 1.00E+15 | 51.0 | 84.2 | 1 | 42.1 | 25.5 | 16.6 |
| 3 | 1.00E+13 | 31.0 | 04.2 | 2 | 42.1 | 25.5 | 16.6 |
| 6 | 1.20E+15 | 61.2 | 101.0 | 1 | 50.5 | 30.6 | 19.9 |
| 0 | 1.20E+15 | 01.2 | 101.0 | 2 | 50.5 | 30.6 | 19.9 |
| 7 | 1.40E+15 | 71.4 | 117.9 | 1 | 59.0 | 35.7 | 23.3 |
| / | | /1.4 | 117.9 | 2 | 58.9 | 35.7 | 23.2 |
| | 1.60E+15 | 81.6 | 134.7 | 1 | 44.9 | 27.2 | 17.7 |
| 8 | | | | 2 | 44.9 | 27.2 | 17.7 |
| | | | | 3 | 44.9 | 27.2 | 17.7 |
| | | | | 1 | 50.5 | 30.6 | 19.9 |
| 9 | 1.80E+15 | 91.8 | 151.5 | 2 | 50.5 | 30.6 | 19.9 |
| | | | | 3 | 50.5 | 30.6 | 19.9 |
| | | | | 1 | 56.2 | 34.0 | 22.2 |
| 10 | 2.00E+15 | 102.0 | 168.4 | 2 | 56.1 | 34.0 | 22.1 |
| | | | | 3 | 56.1 | 34.0 | 22.1 |

| High Dose (3.3e14 vg/kg) | | | | | | | |
|---|---|---|---|---|---|---|---|
| Weight (kg) | Total Dose<br>(vg) | Vector Volume<br>(mL) | Total Volume (mL) | Syringe # | Syringe Volume (mL) | Vector Volume<br>(mL) | Saline Volume<br>(mL) |
| 4 | 1.32E+15 | 67.3 | 67.3 | 1 | 33.7 | 33.7 | 0 |
| 4 | 1.32E+13 | 67.3 | 67.3 | 2 | 33.7 | 33.7 | 0 |
| 5 | 1.65E+15 | 84.2 | 94.3 | 1 | 42.1 | 42.1 | 0 |
| 3 | 1.03E+13 | 84.2 | 84.2 | 2 | 42.1 | 42.1 | 0 |
| ( | 1.00E+15 | 101.0 | 101.0 | 1 | 50.5 | 50.5 | 0 |
| 6 | 1.98E+15 | 101.0 | 101.0 | 2 | 50.5 | 50.5 | 0 |
| 7 | 2.31E+15 | 117.0 | 117.0 | 1 | 58.9 | 58.9 | 0 |
| 7 | | 117.9 | 117.9 | 2 | 58.9 | 58.9 | 0 |
| | 2.64E+15 | 134.7 | | 1 | 44.9 | 44.9 | 0 |
| 8 | | | 134.7 | 2 | 44.9 | 44.9 | 0 |
| | | | | 3 | 44.9 | 44.9 | 0 |
| | | | | 1 | 50.5 | 50.5 | 0 |
| 9 | 2.97E+15 | 151.5 | 151.5 | 2 | 50.5 | 50.5 | 0 |
| | | | | 3 | 50.5 | 50.5 | 0 |
| | | | | 1 | 56.1 | 56.1 | 0 |
| 10 | 3.3E+15 | 168.4 | 168.4 | 2 | 56.1 | 56.1 | 0 |
| | | | | 3 | 56.1 | 56.1 | 0 |

In general, the high dose will not be diluted for a total dose of  $3.3 \times 10^{14} \text{ vg/kg}$ . The low doses will be diluted to the same volume as the high dose and split equally. Thus, the vector will be withdrawn from each vial for the low doses, pooled together, and diluted in an amount of normosol-R to equal the total volume used in the high dose cohort in a given weight range for a total dose of  $6.7 \times 10^{13} \text{ vg/kg}$ .

Preparation of the vector will be done aseptically in a class II BSC by the research staff according to the Manual of Operating Procedures. The vector will be allowed to warm to room temperature prior to infusion to avoid the possibility of particle aggregation following product thaw. The vector-containing syringes will be delivered to the designated PICU suite at NCH. It will be delivered inside a sealed leak-proof bag, carried in a designated container at room temperature and administered to the subject within 8 hours from removal from the -80°C freezer.

# 10.5 Administration

The gene transfer infusion procedure will be performed under sterile conditions in a PICU patient room. The final formulated vector will be administered at 10–20 mL/kg and slowly infused for approximately 60 minutes. Patient-specific dosage based on patient weight recorded during hospital admission on Day -1 will be provided by the pharmacy on procedure date.

## 10.6 Dose Escalation

There will be at least a 3 week intra-cohort dosing interval between dosing of subjects within a cohort to allow review of the safety analysis from five time points (days 1, 2, 7, 14, and 21) prior to dosing of the next subject. There will be at least a 4 week inter-cohort dosing interval

between dosing of subjects in each cohort to allow time for review of the safety analysis of at least six time points (days 1, 2, 7, 14, 21, and 30) from all the subjects within a cohort. Safety analysis will be done by the investigators and the DSMB, as well as, time for decisions to be made about whether to implement a higher dose group. Dose escalation will be based on dose-limiting toxicity (DLT) as described in Section 11.1.1.

The investigators will confer with the IRB and DSMB on all Grade III or higher adverse events with 48 hours that are unanticipated and possibly, probably, or definitely related to the study agent before continuing enrollment. Based on the outcome of the safety and efficacy analysis at the end of each cohort decisions will be made to proceed with dose escalation for the following cohort.

# 10.7 Study Drug Accountability

Upon withdrawal of a vial, the Investigational Product Accountability Log will be recorded with the specific lot number and code of the reagent.

# 10.8 Study Drug Handling and Disposal

Handling of scAAV9.CB.SMN gene will follow compliance standards for Biosafety level 1 vectors following the NIH guidelines. Individuals manipulating the vector will be required to wear adequate personal protective equipment.

All materials used for injection, including sterile drapes, needles, and syringes in contact with the vector will be sealed in leak-proof primary and secondary containers. All waste will be double bagged in autoclave bags bearing the biohazard symbol and sealed with autoclave tape. The bag will then be autoclaved and disposed of in a biohazard waste container.

The empty syringes used for delivery of the vector will be resealed in the procedure room and placed into a small labeled box. The empty vials used to prepare the syringes will also be maintained in the pharmacy. Both will be returned to a secure -80°C freezer archival storage separate from the unused vector storage.

# 11 ASSESSMENTS

## 11.1 Safety Parameters

The primary outcome for this clinical trial is safety. Withdrawal criteria are based on the development of unacceptable toxicity, defined as the occurrence of any one Grade III or higher treatment-related toxicity.

# 11.1.1 Dose Limiting Toxicity

Dose limiting toxicity is defined as any adverse event that is possibly, probably, or definitely related to the study agent. This would include any grade III event, according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03; these classifications are outlined in Table 9.
**Table 9** Adverse Event Classification

| 1 | Mild adverse event; did not require treatment |
|---|---|
| 2 | Moderate adverse event; resolved with treatment |
| 3 | Severe adverse event; inability to carry on normal activities; required professional medical attention |
| 4 | Life-threatening or permanently disabling adverse event |
| 5 | Fatal adverse event |

Study enrollment will be halted by the investigators when any subject experiences a **Grade III**, **or higher** adverse event toxicity that is **unanticipated and possibly**, **probably**, **or definitely related** to the study drug. The event will then be reviewed by the Data Safety Monitoring Board (DSMB) and an evaluation will be made as to whether the trial should be terminated early following the Discontinuation Rules.

#### 11.1.2 Discontinuation Rules

An independent Data Safety Monitoring Board (DSMB) and safety monitor will monitor safety data on a continual basis throughout the trial. The DSMB can recommend early termination of the trial for reasons of safety. Study enrollment will be halted by the investigators when any subject experiences a **Grade III**, **or higher** adverse event toxicity that is **unanticipated and possibly**, **probably**, **or definitely related** to the study drug that presents with clinical symptoms and requires medical treatment. This will include any patient death, important clinical laboratory finding, or any severe local complication in the injected area related to administration of the study agent. If after review by the DSMB, IRB, IBCSC, NIH-OBA and FDA, the decision is made to continue, the study will proceed according to Section 10.6 of this protocol.

# 11.2 Demographic/Medical History

Patient demographics and medical history information will be collected at baseline and captured in the CRF.

#### 11.3 Vital Signs

Vital signs will include blood pressure, respiratory rate, pulse, and axillary temperature at the time points specified in Table 6.

# 11.4 Pulse Oximetry

Pulse oximetry will be measured through a small infrared light attached to the end of the patient's finger.

#### 11.5 Weight and Height

Weight and height will be measured as per the time points specified in Table 6.

# 11.6 Physical Examination

Physical examination will include review of the following systems: HEENT, lungs/thorax, cardiovascular, abdomen, musculoskeletal, neurologic, and genitourinary.

#### 11.7 Vaccination Recommendations

Patients are encouraged to follow all routinely scheduled immunizations as recommended by the Center for Disease Control (CDC). We also recommend seasonal vaccinations that include palivizumab prophylaxis (also known as Synagis) to prevent respiratory syncytial virus (RSV) infections.

### 11.8 Physical Therapy Assessments

#### 11.8.1 CHOP-INTEND

CHOP-INTEND including head control, righting reactions, and trunk movements in supported sitting, supine, and prone positions. Anti-gravity movements in assisted rolling, ventral suspension, and supported standing are also measured. See Appendix 3.

At such time that a subject achieves two consecutive CHOP-INTEND scores of ≥62, a teleconference will be conducted between PI, physical therapist, and AveXis, Inc. to review the subject status and determine whether or not continued CHOP-INTEND assessments are necessary. A decision will be reached and confirmed in writing following the teleconference. If decided that no further assessments are necessary, the physical therapist will cease completion of the CHOP-INTEND assessment at subsequent visits; otherwise CHOP-INTEND assessments will continue monthly.

CHOP-INTEND examinations will be videotaped in accord with the Videotaping Manual.

#### 11.8.2 Bayley Scale of Infant Development version 3

Bayley Scales of Infant Development version 3 is a standardized, norm-referenced infant assessment. The gross and fine motor portions as well as the cognition portion of this test will be administered if the child reaches or exceeds a score of 60 out of 64 on the CHOP-INTEND. The gross and fine motor portion will be completed monthly during the first year and the cognition portion will be completed every three months. During the second year all required portions of the Bayley Scale will be conducted every three months, except for subjects still being seen monthly for CHOP-INTEND assessments. For those subjects the gross and fine motor and cognition portions will be administered as in Year 1. See Appendix 4.

Bayley scales examinations will be videotaped in accord with the Videotaping Manual.

# 11.9 Development Milestones Checklists

The age at which significant motor milestones are achieved will be assessed using a standard Motor Milestone Development Survey shown in Table 10 and a Gross Motor Skills Checklist show in Appendix 5. The Gross Motor Skills Checklist was designed by physical therapists at Nationwide Children's Hospital specifically to assess SMA Type 1 subjects in this trial; it is source from a collection of existing motor assessments.

Additionally, CHOP-INTEND and Bayley physical therapy assessment videos may be transferred to a centralized reviewer for independent determination of milestones achieved.

Table 10 Motor Milestone Development Survey

| 4 months | Prone: Holds head up to vertical axis and legs extended |
|----------|---------------------------------------------------------|
| 6 months | Supine: Rolls over back to front |
| 9 months | Sits alone, with back straight |

| 12 months | Cruises, holding on and may stand without help |
|---|---|
| 15 months | Walks independently |
| 18 months | Runs, walks down stairs one hand held |
| 24 months | Up and down stairs, one step at a time; jumps both feet off floor |
| 30 months | Reciprocal stair climbing; stands on one foot |
| 36 months | Reciprocal stairs going down; rides tricycle |
| 48 months | Hops on one foot; throws ball overhand |
| 60 months | Able to skip |

#### 11.10 Video Evidence

Physical therapy assessments and physician physical examinations required at each study visit will be videotaped in an effort to produce compelling, demonstrable, documented evidence of efficacy, as determined by changes in functional abilities. Parent(s)/legal guardian(s) may also share home videos demonstrating achievement of functional abilities. AveXis, Inc. will provide a secure and confidential upload process for transfer and storage of the videos from NCH to a contracted third-party vendor that will compile and arrange videos as per AveXis, Inc. submission requirements. Any/all videos received at AveXis, Inc. or the contracted vendor will be treated as confidential study data and will be the sole property of AveXis, Inc. AveXis, Inc. and the contracted vendor will provide this secure, encrypted transfer and storage solution to properly protect the identities of patients/families on the videos, which may be shared with regulatory agencies and/or the medical community.

Videos will be provided in a blinded fashion to an independent, centralized reviewer for unbiased assessment of milestone achievement.

#### 11.11 ACTIVE-mini

ACTIVE-mini will be conducted to evaluate infant movement ability. This assessment utilizes the Microsoft Kinect camera interface to capture infant movement with an inexpensive, commercially available camera system with real-time quantitative data output provided. Using the 3 cameras built into the Kinect video, depth and color data of an infant's movement is recorded and analyzed. The Kinect's ability to capture images and simultaneously the distance to every point in each image, provides significantly more information for an assessment of infants, than are captured by current post-processed video-based computer vision systems.

#### 11.12 Electrophysiology Assessments

#### 11.12.1 EIM

Pathological status of muscles will be quantified by EIM. Skulpt, Inc., has developed a handheld device specifically for performing EIM measurements in infants. This device will be used to measure EIM in this study. The device is not yet approved by FDA, but has been tested in over 30 other individuals with no adverse events (AEs) (serious or otherwise) reported to date and currently being tested in SMA infants as part of the Network for Excellence in Neuroscience Clinical Trials (NeuroNEXT) trials. The device has undergone independent electrical safety testing by Intertek (www.intertek.com) to the requirements contained in the following standards:

• IEC 60601-1 Issue 1998/12/01 Ed: 2 Medical Electrical Equipment Part 1: General Requirements and Safety; [Amd. 1-1991(CENELEC EN 60601-1: 1990) (Amd. 2- 1995) (Corrigendum-1995)]

#### 11.12.2 CMAP

The compound muscle action potential (CMAP) size is found using supramaximal stimulation of the motor nerve to the muscle or muscle group (similar to a nerve conduction study). It is recorded using surface electrodes. This is representative of the sum of the surface detected motor unit action potentials from muscles innervated by that nerve.

#### 11.12.3 MUNE

Motor Unit Number Estimation (MUNE) is a technique that uses electromyography to estimate the number of motor units in a muscle. MUNE uses a general formula of:

 $Number\ of\ motor\ units = \frac{compound\ muscle\ action\ potential\ size}{mean\ surface-detected\ motor\ unit\ action\ potential\ size}$ 

#### 11.13 Chest X-ray

A chest x-ray will be performed at screening/baseline.

# 11.14 Swallowing Test

A swallowing test will be performed to determine if the patient has signs of aspiration. If the test is positive for aspiration the patient may be instructed to use an alternative method to oral feeding for the duration of the trial.

#### 11.15 Echocardiography

An ECHO will be performed at screening/baseline and other time points as specified in Table 6.

#### 11.16 Electrocardiogram (ECG)

An ECG will be performed at screening/baseline and other time points as specified in Table 6.

#### 11.17 Pulmonary Assessment

Patients will be assessed by a pulmonologist and may be fitted with a non-invasive positive pressure ventilator (BiPAP) at the discretion of the investigator or study staff.

As part of the pulmonary assessment the parent(s)/legal guardian(s) will be asked by the pulmonologist to recall and report the number of hours per day the subject required ventilation support (including BiPAP) over the two weeks prior to the visit. The response will be recorded in the source documentation.

#### 11.18 Photographs of Infusion Site

Photographs will be taken of the infusion site at the time points specified in Table 6. AveXis, Inc. will provide a secure and confidential upload process for transfer and storage of the photographs from NCH to a contracted third-party vendor that will compile and arrange photographs as per AveXis, Inc. submission requirements. Any/all photographs received at AveXis, Inc. or the contracted vendor will be treated as confidential study data and will be the sole property of AveXis, Inc. AveXis, Inc. and the contracted vendor will provide this secure,

encrypted transfer and storage solution to properly protect the identities of patients/families in the photographs, which may be shared with regulatory agencies and/or the medical community.

## 11.19 Laboratory Assessments

Biological samples will be collected throughout the trial at the time points specified in Table 6.

Laboratory tests with values within the clinically significant range will be repeated during the same visit whenever possible. If the test result returns after the subject leaves the clinic, they will be immediately contacted. Local residents may be asked to return to the outpatient clinic for a repeat test. For non-local residents, arrangements will be made to have the blood test redrawn in a laboratory close to home or by their primary care physician.

**Table 11** Total Blood Volume

| Visit | Tests | Total Volume |
|------------------|----------------------------------------|--------------|
| Screening | Safety, immunology, research | 20 mL |
| Day 0 | Safety, immunology | 15 mL |
| Day 7 | Safety, immunology | 15 mL |
| Day 14 | Safety, immunology | 15 mL |
| Day 21 | Safety, immunology, research | 20 mL |
| Day 30 | Safety, immunology, research | 20 mL |
| Day 60 | Safety, immunology, research | 20 mL |
| Day 90 | Safety, immunology, research | 20 mL |
| Day 180 | Safety, immunology, research | 20 mL |
| Day 270 | Safety, immunology, research | 20 mL |
| Day 360 | Safety, immunology, research | 20 mL |
| Day 450 | Safety, immunology, research | 20 mL |
| Day 540 | Safety, immunology, research | 20 mL |
| Day 630 | Safety, immunology, research | 20 mL |
| Last Study Visit | Safety, immunology, research | 20 mL |
| | Total Volume for Study 2-Year Duration | 285 mL |

In a case where sufficient blood cannot be collected from a patient, blood will be used in the following priority order with the first having greatest priority and last having the least priority:

- 1. Safety blood labs
- 2. Serum antibody to AAV9
- 3. IFN-y ELISpots to detect T-cell responses
- 4. Research Blood sample stored for future purposes

#### 11.19.1 Hematology

Hematology analysis will include a CBC with differential and platelet with smear.

# 11.19.2 Blood Chemistry

Chemistry analysis will include the following at all study visits:

- serum GGT
- AST/ALT
- serum total bilirubin
- direct bilirubin
- albumin
- glucose
- total creatine kinase and iso-enzyme (CK-MB)
- troponin
- creatinine/BUN
- electrolytes
- alkaline phosphatase
- amylase

Study Visit 2 will also include:

• serum protein electrophoresis (SPEP)

# 11.19.3 Urinalysis

Urine samples will be collected via cotton swabs. Urinalysis will include the following parameters:

- Color
- Clarity/turbidity
- pH
- Specific gravity
- Glucose
- Ketones
- Nitrites
- Leukocyte esterase
- Bilirubin
- Urobilirubin
- Blood
- Protein
- RBCs
- WBCs
- Squamous epithelial cells

Casts

- Crystals
- Bacteria
- Yeast

#### 11.19.4 Coagulation Studies

Coagulation studies including prothrombin time (PT), PTT, and INR will be performed at the time points specified in Table 6.

## 11.19.5 Capillary Blood Gas

A puncture or small incision will be made with a lancet or similar device into the cutaneous layer of the patient's skin at a highly vascularized area (heel, finger, toe). To accelerate blood flow and reduce the difference between the arterial and venous gas pressures, the area will be warmed prior to the puncture. As the blood flows freely from the puncture site, the sample will be collected in a heparinized glass capillary tube.

### 11.19.6 Virus Serology

Patients will be tested for HIV and have a serology test for hepatitis B and C.

# 11.19.7 Research Immunology Blood

Blood samples will be collected to test for serum antibodies to AAV9 and SMN.

# 11.19.8 Baseline Screening of Mother

There is a potential that the mother of the enrolled infant may have pre-existing antibodies to AAV9 that may be transferred to the patient through breast milk or theoretically via placental transfer in utero. Informed consent will be requested from the mother of the infant to screen the mother for circulating antibodies to AAV9. Once informed consent has been obtained, the mother will have her blood drawn from a peripheral vein for screening of anti-AAV9 antibodies.

#### 11.19.9 IFN-y ELISpots

Blood will be collected to perform IFN- $\gamma$  ELISpots to detect T-cell responses to AAV9 and SMN.

#### 11.19.10 Research Blood Sample

Blood samples will be collected for future research purposes, to examine/research potential disease modifiers and/or biomarkers. Research blood will also be used for exon 7 modifier testing at screening. Additionally, blood samples collected for research may be transferred to an independent third-party laboratory contracted by AveXis, Inc. such that genetic testing confirming SMA Type 1 diagnosis can be re-confirmed for each subject.

An additional blood sample may be collected and provided to an independent laboratory for reconfirmatory genetic testing.

#### 11.19.11 Saliva, Urine, and Stool Collection

Saliva, urine, and stool samples will be collected for viral shedding studies. Saliva will be collected from the patient's mouth with a pipette and oral swab.  $200\text{-}500~\mu\text{L}$  of urine will be collected from patients' soiled diapers by soaking a cotton ball. Pea-sized fecal samples will be collected from patients' soiled diapers. Each of these samples will be placed in a

DNAse/RNAse-free Eppendorf tube with locking top. The tubes will be stored in a -80°C freezer.

#### 12 ADVERSE AND SERIOUS ADVERSE EVENTS

#### 12.1 Definition of Adverse Events

### 12.1.1 Adverse Event (AE)

An AE is the development of an undesirable medical condition or the deterioration of a preexisting medical condition following or during exposure to a pharmaceutical product, whether or not considered casually related to the product. In clinical studies, an AE can include an undesirable medical condition occurring at any time, including baseline or washout periods, even if no study treatment has been administered.

All AEs that occur after any patient has been enrolled, before treatment, during treatment, or within 30 days of the last study visit, whether or not they are related to the study, must be recorded in the eCRF.

#### 12.1.2 Serious Adverse Event (SAE)

A serious adverse event is an AE occurring during any study phase (i.e., baseline, treatment, washout, or follow-up), and at any dose of the investigational product, comparator or placebo, that fulfils one or more of the following:

- Results in death
- It is immediately life-threatening
- It requires in-patient hospitalization or prolongation of existing hospitalization
- It results in persistent or significant disability or incapacity
- Results in a congenital abnormality or birth defect
- It is an important medical event that may jeopardize the patient or may require medical intervention to prevent one of the outcomes listed above.

All SAEs that occur after any patient has signed informed consent, before treatment, during treatment, or within 30 days following the last study visit, whether or not they are related to the study, must be recorded on forms provided by AveXis, Inc.

#### 12.1.3 Other Adverse Event (OAE)

OAEs may be identified by the Drug Safety Physician and, if applicable, also by the Clinical Study Team Physician during the evaluation of safety data for the Clinical Study Report. Significant adverse events of particular clinical importance, other than SAEs and those AEs leading to discontinuation of the patient/subject from the study, will be classified as OAEs. For each OAE, a narrative may be written and included in the Clinical Study Report.

#### 12.2 Relationship to Study Drug

An Investigator who is qualified in medicine must make the determination of relationship to the investigational product for each AE (Unrelated, Possibly Related or Probably Related). The Investigator should decide whether, in his or her medical judgment, there is a reasonable possibility that the event may have been caused by the investigational product. If no valid reason

exists for suggesting a relationship, then the AE should be classified as "unrelated." If there is any valid reason, even if undetermined, for suspecting a possible cause-and-effect relationship between the investigational product and the occurrence of the AE, then the AE should be considered "related."

If the relationship between the AE/SAE and the investigational product is determined to be "possible" or "probable" the event will be considered to be related to the investigational product for the purposes of expedited regulatory reporting.

# 12.3 Recording Adverse Events

Adverse events spontaneously reported by the patient and/or in response to an open question from the study personnel or revealed by observation will be recorded during the study at the investigational site. Clinically significant changes in laboratory values, blood pressure, and pulse need not be reported as AEs. However, abnormal values that constitute an SAE or lead to discontinuation of administration of study drug must be reported and recorded as an AE. Information about AEs will be collected from Day -1 until the end of the study. Serious Adverse Event information will be collected from signing of the consent form until 30 days following the last study visit. The AE term should be reported in standard medical terminology when possible. For each AE, the investigator will evaluate and report the onset (date and time), resolution (date and time), intensity, causality, action taken, serious outcome (if applicable), and whether or not it caused the patient to discontinue the study.

Events will be graded in accord with Table 9.

It is important to distinguish between serious and severe AEs. Severity is a measure of intensity whereas seriousness is defined by the criteria under Section 12.1.2. An AE of severe intensity may not be considered serious.

#### 12.4 Reporting Adverse Events

All SAEs (related and unrelated) will be recorded from the signing of consent form until 30 days following the last study visit. Any SAEs considered possibly or probably related to the investigational product and discovered by the Investigator at any time after the study should be reported. All SAEs must be reported to AveXis, Inc. within 24 hours of the first awareness of the event. The Investigator must complete, sign and date the SAE pages, verify the accuracy of the information recorded on the SAE pages with the corresponding source documents, and send notification to AveXis, Inc., as per the Safety Management Plan.

Additional follow-up information, if required or available, should all be provided to AveXis, Inc. within 5 calendar days of receipt for events that are unexpected and/or possibly/probably/definitely related to the investigational product. This information should be provided on a follow-up SAE form and placed with the original SAE information and kept with the appropriate section of the eCRF and/or study file. Follow-up information for events that are not unexpected and are not related to the investigational product should be provided to AveXis, Inc. within 7 calendar days of receipt.

AveXis, Inc. is responsible for notifying the relevant regulatory authorities of certain events. It is the Principal Investigator's responsibility to notify the IRB of all SAEs that occur at his or her site, as per the IRB's reporting guidelines.

AveXis, Inc. will review the safety database at least quarterly; this data will also be provided to the DSMB for quarterly review. If AveXis or the DSMB determines there are any emerging safety signals and/or trends that may warrant reporting to appropriate regulatory authorities, AveXis will report these events in aggregate.

#### 13 DATA SAFETY MONITORING BOARD

The Data and Safety Monitoring Board (DSMB) will act in an advisory capacity to review participant safety and study progress for the clinical trial. Responsibilities of the DSMB are to:

- review the research protocol, informed consent documents and plans for data and safety monitoring;
- evaluate the progress of the trial, including periodic assessments of data quality and timeliness, participant recruitment, accrual and retention, participant risk versus benefit, trial site performance, and other factors that can affect study outcome;
- consider factors external to the study when relevant information becomes available, such as scientific or therapeutic developments that may have an impact on participant safety or the ethics of the trial;
- review study performance, make recommendations and assist in the resolution of problems reported by the Principal Investigator;
- protect the safety of the study participants;
- review safety data to determine whether to recommend dose escalation;
- review quarterly safety data to determine safety signals or trends;
- ensure the confidentiality of the trial data and the results of monitoring; and,
- assist by commenting on any problems with study conduct, enrollment, and sample size and/or data collection.

#### 13.1 DSMB Reporting and Meetings

Reports describing the status of the study will be prepared by AveXis, Inc. and/or the Principal Investigator's staff and sent to the DSMB at least quarterly, or at the DSMB's request. A meeting (either by teleconference or webcast) with the DSMB will be scheduled after Day 30 visit of the last patient in each cohort, or at the DSMB's request. Reports will be submitted prior to a scheduled meeting for review by the DSMB.

Reports will include the following:

- A brief narrative of the study status, including the target enrollment, current and projected time to completing enrollment. Any significant events and/or difficulties should be briefly described in this narrative;
- A brief narrative for each participant describing gender, age, race and ethnicity and other relevant demographic characteristics. The narrative for each participant should briefly describe his/her study status (i.e., dose level, visit number, adverse event information);

• A timeline outlining the study progress relative to visit number for each participant, as well as time points for each SAE/Dose Limiting Toxicity. A total for Adverse Events (AEs) for each participant should be included;

- A summary of AEs by classification;
- A listing of AE details grouped by participant;
- A listing of SAE details grouped by participant;
- A listing of deaths;
- A summary of clinically significant laboratory test results;
- A listing of protocol deviations.

# 13.2 DSMB Membership

The DSMB membership will consist of persons completely independent of the investigator and sponsor who have no financial, scientific, or other conflicts of interest with the trial. Current or past collaborators or associates of Dr. Mendell or AveXis, Inc. must note any conflict of interest before their eligibility to serve on the DSMB is approved. The DSMB will include experts in or representatives of the fields of:

- Neurology and Neuromuscular Diseases
- Immunology
- Gene Therapy
- Spinal Muscular Atrophy Clinical Care
- Clinical Research and Clinical Trials
- Statistics (non-voting member)

Individuals invited to serve on the DSMB as either voting or non-voting members must disclose any potential conflicts of interest, whether real or perceived. Conflicts of interest can include professional, proprietary, and miscellaneous interests as described in 45 CFR Part 94. Potential conflicts that develop during a member's tenure on a DSMB must also be disclosed. Written documentation attesting to an absence of conflict of interest is required annually.

AveXis, Inc. will employ a third party to provide planning, organization, preparation, and oversight services for the DSMB meetings.

#### 14 STATISTICS

This is a Phase I trial, with safety as the primary measure. A secondary outcome includes the time to death or  $\geq 16$ -hour respiratory assistance per day continuously for  $\geq 2$  weeks in the absence of an acute reversible illness. Only patients with 2 copies of SMN2 will be enrolled. 92% of SMA Type 1 patients with two copies of SMN2 live  $\leq 21$  months. For this study the primary end point for efficacy will be death or  $\geq 16$  hour respiratory assistance per day (includes BiPAP). A successful measure for efficacy for this study will be 50% of SMA Type 1 subjects living with less than 16 hour respiratory assistance at 2 years of age.

#### 15 DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

#### 15.1 Study Monitoring

During the study, a monitor from AveXis, Inc. or representative will have regular contact with the investigational site, for the following:

- Provide information and support to the investigator(s)
- Confirm that facilities remain acceptable
- Confirm that the investigational team is adhering to the protocol and ICH/GCP guidelines, that data are being accurately recorded in the case report forms, and that investigational product accountability checks are being performed
- Perform source data verification. This includes a comparison of the data in the case report forms with the patient's medical records at the hospital or practice, and other records relevant to the study. This will require direct access to all original records for each patient (e.g., clinic charts) including access to the site's Electronic Medical Record (EMR) and the videos captured during specified visit assessments.
- Record and report any protocol deviations not previously sent to AveXis, Inc.
- Confirm AEs and SAEs have been properly documented on eCRFs and confirm any SAEs have been forwarded to AveXis, Inc. and those SAEs that met criteria for reporting have been forwarded to the IRB.

The monitor will be available between visits if the investigator(s) or other staff needs information or advice.

#### 15.2 Audits and Inspections

Authorized representatives of AveXis, Inc., a regulatory authority, or an Institutional Review Board may visit the site to perform audits or inspections, including source data verification. The purpose of an AveXis, Inc. audit or inspection is to systematically and independently examine all study-related activities and documents to determine whether these activities were conducted, and data were recorded, analyzed, and accurately reported according to the protocol, Good Clinical Practice guidelines of the International Conference on Harmonization, and any applicable regulatory requirements. The investigator should contact AveXis, Inc. immediately if contacted by a regulatory agency about an inspection.

### 15.3 Institutional Review Board (IRB)

The Principal Investigator must obtain IRB approval for the investigation. Initial IRB approval, and all materials approved by the IRB for this study including the patient consent form and recruitment materials must be maintained by the Investigator and made available for inspection.

# 15.4 Quality Control and Quality Assurance

To ensure compliance with Good Clinical Practices and all applicable regulatory requirements, AveXis, Inc. may conduct a quality assurance audit. Please see Section 15.2 for more details regarding the audit process.

#### 16 ETHICS

#### 16.1 Ethics Review

The final study protocol, including the final version of the Informed Consent Form, must be approved or given a favorable opinion in writing by an IRB or IEC as appropriate.

The Principal Investigator is responsible for informing the IRB of any amendment to the protocol in accordance with local requirements. The protocol must be re-approved by the IRB upon receipt of amendments and annually, as local regulations require.

The Principal Investigator is also responsible for providing the IRB with reports of any reportable serious adverse drug reactions from any other study conducted with the investigational product. AveXis, Inc. will provide this information to the Principal Investigator.

Progress reports and notifications of serious adverse drug reactions will be provided to the IRB according to local regulations and guidelines.

#### 16.2 Ethical Conduct of the Study

The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki (Appendix 1) and are consistent with ICH/Good Clinical Practice, applicable regulatory requirements and AveXis, Inc.'s policy on Bioethics.

#### 16.3 Written Informed Consent

The Principal Investigator(s) will ensure that the patient is given full and adequate oral and written information about the nature, purpose, possible risk and benefit of the study. Patients must also be notified that they are free to discontinue from the study at any time. The patient should be given the opportunity to ask questions and allowed time to consider the information provided.

The patient's signed and dated informed consent must be obtained before conducting any study procedures.

The Principal Investigator(s) must maintain the original, signed Informed Consent Form. A copy of the signed Informed Consent Form must be given to the patient.

Per the National Institutes of Health's Guidelines for Research Involving Recombinant or Synthetic Nucleic Acid Molecules (http://oba.od.nih.gov), an autopsy must be requested should a study participant die following participation in a gene transfer trial, no matter what the cause of death. An autopsy is requested to obtain vital information about the safety and efficacy of gene transfer. Patients' parent(s)/legal guardians will be asked to provide consent for an autopsy in advance of any death. Consent is requested at the beginning of the study to relieve the burden of making such a decision at the time of death should such a terrible and unfortunate event occur.

# 17 DATA HANDLING AND RECORDKEEPING

# 17.1 Electronic Case Report Forms

Adequate and accurate case records will be maintained and all relevant observations and data related to the study will be recorded. This will include medical history/ physical examination, hematology, clinical chemistry and serology results, a check list of inclusion and exclusion

criteria, urinary screening, drug administration, and a record of sample collection, hemodynamic measurements, clinical assessments, AEs, and final evaluation.

Electronic CRFs will be used in this study. The eCRF will be electronically signed and dated by the Principal Investigator or his designee after his/her review. After the completion of the study, completed eCRFs will be retained in the archives.

Completed eCRFs will be reviewed by the study monitor against the source documentation for accuracy and completeness. Once signed by the Investigator, the monitor will transmit the completed eCRFs to data management for data validation and database analysis.

### 17.2 Inspection of Records

AveXis, Inc. will be allowed to conduct site visits to the investigation facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the monitor to inspect the drug storage area, study drug stocks, drug accountability records, subject charts, study source documents, and other records relative to study conduct.

#### 17.3 Retention of Records

All primary data that are a result of the original observations and activities of the study and that are necessary for the reconstruction and evaluation of any study report will be retained in a secure archive at the study site for a period not less than 2 years after the last approval of a marketing application in an ICH region, and until there are no pending or contemplated marketing applications in an ICH region, or until at least 2 years have lapsed since the formal discontinuation of the clinical development of the investigational product.

The site will maintain a Clinical Study Document Binder, which will be maintained at the study site. In this binder, there will be tabbed sections for study documents including the following: study personnel identification and signature list, subject screening records, subject roster (names omitted), protocol and amendments or administrative changes, FDA Form 1572 (if required), study staff Curricula Vitae, IRB documentation, an approved sample ICF, drug accountability records, correspondence, site monitoring reports, blank Data Documentation form, and lab accreditations and normal values. The site must keep this binder current and available for review by the Sponsor, IRB, and/or FDA.

# 17.4 Retention of Samples

The identified storage laboratory will be responsible for arranging storage of any remaining or unused biological samples as well as properly documenting the storage procedures, once all study-required analyses are complete, as per sample processing requirements until such time that AveXis, Inc. provides external storage vendor transfer or destruction instructions.

#### 18 PUBLICATION POLICY

The investigator is obliged to provide the Sponsor with complete test results and all data derived by the investigator from the study. During the study, only the Sponsor may make study information available to other study investigators or to regulatory agencies, except as required by law or regulation or as otherwise agreed upon in writing by Sponsor and investigator. Except as otherwise allowable in the clinical study site agreement, any public disclosure (including publicly accessible websites) related to the protocol or study results, other than study recruitment materials and/or advertisements, is the sole responsibility of the Sponsor.

Manuscript authorship for any peer-reviewed publication will appropriately reflect contributions to the production and review of the document (in accordance with ICJME). All publications and presentations must be prepared in accordance with this section and the Clinical Study Site Agreement. In the event of any discrepancy between the protocol and the Clinical Study Site Agreement, the Clinical Study Site Agreement will prevail.

The investigator will provide the Sponsor with a copy of any proposed publication or presentation for review and comment at least 30 days prior to such presentation or submission for publication. The Sponsor shall inform the investigator in writing of any changes or deletions in such presentation or publication required to protect the Sponsor's confidential and proprietary technical information and to address inaccurate data or inappropriate interpretations in the context of any pooled multicenter results. At the expiration of such 30-day period, the investigator may proceed with the presentation or submission for publication unless the Sponsor has notified the institution or the investigator in writing that such proposed publication or presentation discloses the Sponsor's confidential and proprietary technical information. Further, upon the request of the Sponsor, the investigator will delay the publication or presentation for an additional 60 days to permit the Sponsor to take necessary actions to protect its intellectual property interests. In the event of any discrepancy between the protocol and the Clinical Study Site Agreement, the Clinical Study Site Agreement will prevail.

#### 19 LIST OF REFERENCES

1. Mercuri E, Bertini E, Iannaccone ST. Childhood spinal muscular atrophy: controversies and challenges. *Lancet neurology* 2012; 11(5): 443-52.

- 2. Kolb SJ, Kissel JT. Spinal muscular atrophy: a timely review. *Archives of neurology* 2011; 68(8): 979-84.
- 3. Lefebvre S, Burglen L, Reboullet S, Clermont O, Burlet P, Viollet L *et al.* Identification and characterization of a spinal muscular atrophy-determining gene. *Cell* 1995; 80(1): 155-64.
- 4. Lorson CL, Hahnen E, Androphy EJ, Wirth B. A single nucleotide in the SMN gene regulates splicing and is responsible for spinal muscular atrophy. *Proceedings of the National Academy of Sciences of the United States of America* 1999; 96(11): 6307-11
- 5. Monani UR, Lorson CL, Parsons DW, Prior TW, Androphy EJ, Burghes AH *et al.* A single nucleotide difference that alters splicing patterns distinguishes the SMA gene SMN1 from the copy gene SMN2. *Human molecular genetics* 1999; 8(7): 1177-83.
- 6. Lefebvre S, Burlet P, Liu Q, Bertrandy S, Clermont O, Munnich A *et al.* Correlation between severity and SMN protein level in spinal muscular atrophy. *Nature genetics* 1997; 16(3): 264-9.
- 7. Park GH, Kariya S, Monani UR. Spinal muscular atrophy: new and emerging insights from model mice. *Current neurology and neuroscience reports* 2010; 10(2): 108-17.
- 8. Feldkotter M, Schwarzer V, Wirth R, Wienker TF, Wirth B. Quantitative analyses of SMN1 and SMN2 based on real-time lightCycler PCR: fast and highly reliable carrier testing and prediction of severity of spinal muscular atrophy. *American journal of human genetics* 2002; 70(2): 358-68.
- 9. Farrar MA, Vucic S, Johnston HM, du Sart D, Kiernan MC. Pathophysiological Insights Derived by Natural History and Motor Function of Spinal Muscular Atrophy. *The Journal of pediatrics* 2012.
- 10. Swoboda KJ, Prior TW, Scott CB, McNaught TP, Wride MC, Reyna SP *et al.* Natural history of denervation in SMA: relation to age, SMN2 copy number, and function. *Annals of neurology* 2005; 57(5): 704-12.
- 11. Le TT, McGovern VL, Alwine IE, Wang X, Massoni-Laporte A, Rich MM *et al.* Temporal requirement for high SMN expression in SMA mice. *Human molecular genetics* 2011; 20(18): 3578-91.
- 12. Farrar MA, Vucic S, Johnston HM, Kiernan MC. Corticomotoneuronal integrity and adaptation in spinal muscular atrophy. *Archives of neurology* 2012; 69(4): 467-73.
- 13. Foust KD, Wang X, McGovern VL, Braun L, Bevan AK, Haidet AM *et al.* Rescue of the spinal muscular atrophy phenotype in a mouse model by early postnatal delivery of SMN. *Nature biotechnology* 2010; 28(3): 271-4.
- 14. Sugarman EA, Nagan N, Zhu H, Akmaev VR, Zhou Z, Rohlfs EM *et al.* Pan-ethnic carrier screening and prenatal diagnosis for spinal muscular atrophy: clinical laboratory analysis of >72,400 specimens. *European journal of human genetics : EJHG* 2012; 20(1): 27-32.

15. Riessland M, Ackermann B, Forster A, Jakubik M, Hauke J, Garbes L *et al.* SAHA ameliorates the SMA phenotype in two mouse models for spinal muscular atrophy. *Human molecular genetics* 2010; 19(8): 1492-506.

- 16. Dayangac-Erden D, Bora-Tatar G, Dalkara S, Demir AS, Erdem-Yurter H. Carboxylic acid derivatives of histone deacetylase inhibitors induce full length SMN2 transcripts: a promising target for spinal muscular atrophy therapeutics. *Arch Med Sci* 2011; 7(2): 230-4.
- 17. Darbar IA, Plaggert PG, Resende MB, Zanoteli E, Reed UC. Evaluation of muscle strength and motor abilities in children with type II and III spinal muscle atrophy treated with valproic acid. *BMC Neurol* 2011; 11: 36.
- 18. Butchbach ME, Edwards JD, Burghes AH. Abnormal motor phenotype in the SMNDelta7 mouse model of spinal muscular atrophy. *Neurobiology of disease* 2007; 27(2): 207-19.
- 19. Mendell JR, Rodino-Klapac LR, Rosales-Quintero X, Kota J, Coley BD, Galloway G et al. Limb-girdle muscular dystrophy type 2D gene therapy restores alphasarcoglycan and associated proteins. Annals of neurology 2009; 66(3): 290-7.
- 20. Finkel RS, McDermott MP, Kaufmann P, Darras BT, Chung WK, Sproule DM, Kang PB, Foley AR, Yang ML, Martens WB, Oskoui M, Glanzman AM, Flickinger J, Montes J Dunaway S, O'Hagen J, Quigley J, Riley S, Benton M, Ryan PA, Montgomery M, Marra J, Gooch C, De Vivo DC. Finkel et al 2014: Observational study of spinal muscular atrophy type I and implications for clinical trials. *Neurology*. 2014 Aug 26;83(9):810-7.

#### **20 APPENDICES**

# APPENDIX 1 DECLARATION OF HELSINKI: ETHICAL PRINCIPLES FOR MEDICAL RESEARCH INVOLVING HUMAN SUBJECTS

Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964 and amended by the:

29th WMA General Assembly, Tokyo, Japan, October 1975

35th WMA General Assembly, Venice, Italy, October 1983

41st WMA General Assembly, Hong Kong, September 1989

48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996

52nd WMA General Assembly, Edinburgh, Scotland, October 2000

53rd WMA General Assembly, Washington DC, USA, October 2002 (Note of Clarification added)

55th WMA General Assembly, Tokyo, Japan, October 2004 (Note of Clarification added)

59th WMA General Assembly, Seoul, Republic of Korea, October 2008

64th WMA General Assembly, Fortaleza, Brazil, October 2013

- 1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data.
  - The Declaration is intended to be read as a whole and each of its constituent paragraphs should be applied with consideration of all other relevant paragraphs.
- 2. Consistent with the mandate of the WMA, the Declaration is addressed primarily to physicians. The WMA encourages others who are involved in medical research involving human subjects to adopt these principles.

#### **General Principles**

- 3. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 4. It is the duty of the physician to promote and safeguard the health, well-being and rights of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- 5. Medical progress is based on research that ultimately must include studies involving human subjects.
- 6. The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best proven interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 7. Medical research is subject to ethical standards that promote and ensure respect for all human subjects and protect their health and rights.

8. While the primary purpose of medical research is to generate new knowledge, this goal can never take precedence over the rights and interests of individual research subjects.

- 9. It is the duty of physicians who are involved in medical research to protect the life, health, dignity, integrity, right to self-determination, privacy, and confidentiality of personal information of research subjects. The responsibility for the protection of research subjects must always rest with the physician or other health care professionals and never with the research subjects, even though they have given consent.
- 10. Physicians must consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.
- 11. Medical research should be conducted in a manner that minimizes possible harm to the environment.
- 12. Medical research involving human subjects must be conducted only by individuals with the appropriate ethics and scientific education, training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional.
- 13. Groups that are underrepresented in medical research should be provided appropriate access to participation in research.
- 14. Physicians who combine medical research with medical care should involve their patients in research only to the extent that this is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- 15. Appropriate compensation and treatment for subjects who are harmed as a result of participating in research must be ensured.

#### Risks, Burdens and Benefits

- 16. In medical practice and in medical research, most interventions involve risks and burdens.

  Medical research involving human subjects may only be conducted if the importance of the objective outweighs the risks and burdens to the research subjects.
- 17. All medical research involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and groups involved in the research in comparison with foreseeable benefits to them and to other individuals or groups affected by the condition under investigation.
  - Measures to minimize the risks must be implemented. The risks must be continuously monitored, assessed and documented by the researcher.
- 18. Physicians may not be involved in a research study involving human subjects unless they are confident that the risks have been adequately assessed and can be satisfactorily managed.

When the risks are found to outweigh the potential benefits or when there is conclusive proof of definitive outcomes, physicians must assess whether to continue, modify or immediately stop the study.

#### **Vulnerable Groups and Individuals**

- 19. Some groups and individuals are particularly vulnerable and may have an increased likelihood of being wronged or of incurring additional harm.
  - All vulnerable groups and individuals should receive specifically considered protection.
- 20. Medical research with a vulnerable group is only justified if the research is responsive to the health needs or priorities of this group and the research cannot be carried out in a non-vulnerable group. In addition, this group should stand to benefit from the knowledge, practices or interventions that result from the research.

#### Scientific Requirements and Research Protocols

- 21. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 22. The design and performance of each research study involving human subjects must be clearly described and justified in a research protocol.

The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, potential conflicts of interest, incentives for subjects and information regarding provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study.

In clinical trials, the protocol must also describe appropriate arrangements for post-trial provisions.

#### **Research Ethics Committees**

23. The research protocol must be submitted for consideration, comment, guidance and approval to the concerned research ethics committee before the study begins. This committee must be transparent in its functioning, must be independent of the researcher, the sponsor and any other undue influence and must be duly qualified. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration.

The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No amendment to the protocol may be made without consideration and approval by the committee. After the end of the study, the researchers must submit a final report to the committee containing a summary of the study's findings and conclusions.

#### **Privacy and Confidentiality**

24. Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information.

#### **Informed Consent**

- 25. Participation by individuals capable of giving informed consent as subjects in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no individual capable of giving informed consent may be enrolled in a research study unless he or she freely agrees.
- 26. In medical research involving human subjects capable of giving informed consent, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, post-study provisions and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information.

After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.

All medical research subjects should be given the option of being informed about the general outcome and results of the study.

- 27. When seeking informed consent for participation in a research study the physician must be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent must be sought by an appropriately qualified individual who is completely independent of this relationship.
- 28. For a potential research subject who is incapable of giving informed consent, the physician must seek informed consent from the legally authorized representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the group represented by the potential subject, the research cannot instead be performed with persons capable of providing informed consent, and the research entails only minimal risk and minimal burden.
- 29. When a potential research subject who is deemed incapable of giving informed consent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorized representative. The potential subject's dissent should be respected.
- 30. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research group. In such circumstances the physician must seek informed consent from the legally authorized representative. If no such representative is available and if the research cannot be delayed,

the study may proceed without informed consent provided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research must be obtained as soon as possible from the subject or a legally authorized representative.

- 31. The physician must fully inform the patient which aspects of their care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never adversely affect the patient-physician relationship.
- 32. For medical research using identifiable human material or data, such as research on material or data contained in biobanks or similar repositories, physicians must seek informed consent for its collection, storage and/or reuse. There may be exceptional situations where consent would be impossible or impracticable to obtain for such research. In such situations the research may be done only after consideration and approval of a research ethics committee.

#### Use of Placebo

33. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best proven intervention(s), except in the following circumstances:

Where no proven intervention exists, the use of placebo, or no intervention, is acceptable; or where for compelling and scientifically sound methodological reasons the use of any intervention less effective than the best proven one, the use of placebo, or no intervention is necessary to determine the efficacy or safety of an intervention and the patients who receive any intervention less effective than the best proven one, placebo, or no intervention will not be subject to additional risks of serious or irreversible harm as a result of not receiving the best proven intervention. Extreme care must be taken to avoid abuse of this option.

#### **Post-Trial Provisions**

34. In advance of a clinical trial, sponsors, researchers and host country governments should make provisions for post-trial access for all participants who still need an intervention identified as beneficial in the trial. This information must also be disclosed to participants during the informed consent process.

#### Research Registration and Publication and Dissemination of Results

- 35. Every research study involving human subjects must be registered in a publicly accessible database before recruitment of the first subject.
- 36. Researchers, authors, sponsors, editors and publishers all have ethical obligations with regard to the publication and dissemination of the results of research. Researchers have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. All parties should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results must be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest must be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

# **Unproven Interventions in Clinical Practice**

37. In the treatment of an individual patient, where proven interventions do not exist or other known interventions have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorized representative, may use an unproven intervention if in the physician's judgement it offers hope of saving life, reestablishing health or alleviating suffering. This intervention should subsequently be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information must be recorded and, where appropriate, made publicly available.

#### APPENDIX 2 AUTOPSY PLAN

Regional Pathology and Autopsy Services, Inc., a nationwide company that provides autopsy and tissue collection services, will perform autopsy and tissue collection for the patients in the clinical trial. This company will deploy a pathology assistant to the funeral home of the deceased to perform the autopsy and tissue collection. Standard autopsy incisions are used to perform the autopsy and pathology necessary to determine the cause of death, which will be completed by Regional Pathology and Autopsy Services.

During the procedure, multiple tissues along with the entire spinal cord will be collected for research purposes. Up to 7 sections or pieces from each organ and each region of the spinal cord will be collected and returned to the principal investigator of the trial at Nationwide Children's Hospital. Analysis of the tissue will be done to determine whether the vector transduced the expected motor neurons and if the SMN gene was expressed. These results demonstrate whether the vector delivered the therapeutic gene as expected. Tissue samples collected will also be available for histology and immunohistochemistry, allowing the state of the motor neurons and muscles to be examined.

Specifically, tissue samples from the following organs and regions of the spinal cord and brain will be collected (see Table 12 below). Tissue sample will be frozen or fixed (eg. 2% paraformaldehyde) for appropriate analysis.

Families will be asked to consent to the autopsy and tissue collection prior to any sign of moribund or death by the clinical team conducting the trial. There are distinct consent forms for the formal autopsy and for the research tissue collection. This allows the families the flexibility to participate in one or both of the research activities.

**Table 12** Tissue Samples for Analysis

| Brain | Spinal Cord | Muscles | Organs |
|---|---|---|---|
| Motor cortex | Cervical spinal cord | Diaphragm | Spleen |
| Layer 5 motor cortex | Thoracic<br>spinal cord | #6/#7 Rib<br>with<br>intercostal<br>muscle and<br>nerve | Kidney |
| Brain stem | Lumbar spinal cord | Psoas muscle | Small intestine |
| | Sacral spinal cord | | Large<br>intestine |
| | Dorsal root | | Pancreas |
| | cervical level | | Stomach |
| | Ventral root | | Lung |
| | cervical level | | Heart |
| | DRG root | | Liver |
| | cervical level | | Inguinal<br>Iymph node |
| | Cerebrospinal fluid | | Gonads |

# APPENDIX 3 CHOP-INTEND

# CHILDREN'S HOSPITAL of PHILADELPHIA INFANT TEST OF NEUROMUSCULAR DISORDERS

| Time of evalu | uation: | | (AM/PM) Hours off BiPAP at testing: | | | <u>(h)</u> |
|---|---|---|---|---|---|---|
| Item | Position | Test Procedure | Graded Response | | Score | |
| 1 | Supine | Observe throughout | Antigravity shoulder movement (achieves elbow off surface) | 4 | L | Best side: |
| Spontaneous<br>movement | | <u>testing</u> | Antigravity elbow movement (achieves hand and forearm off surface) | 3 | | |
| (Upper | | May unweight limb or stimulate infant to facilitate response | Wrist movement | 2 | D | State: |
| extremity) | | | Finger movement | Score Best side: | | |
| | | Observe throughout testing May unweight limb or stimulate infant Antigravity hip movement (achieves feet and knees off surface) Antigravity hip adduction/internal rotation (knees off surface) Active gravity eliminated knee movement | | | | |
| 2 | Supine | testing May unweight limb or stimulate infant to facilitate response | Antigravity hip movement (achieves feet and knees off surface) | 4 | L | Best side: |
| Spontaneous<br>movement | | Antigravity hip adduction/internal rotation (knees off surface) | 3 | | | |
| (Lower | (Lawar May unw | | Active gravity eliminated knee movement | 2 | D | State: |
| extremity) | | | Ankle movement | 1 | K | |
| | | No movement of limbs | 0 | | | |
| 3 | Supine | Grip strength: place finger in palm and lift until shoulder comes off surface | Maintains hand grip with shoulder off bed | 4 | L | Best side: |
| Hand grip | | observe when infant loses grasp<br>May use toy of similar diameter for | Maintains grip with elbow off surface (shoulders on surface) | 3 | | |
| | | older children | Maintains grip with forearm off surface (elbow supported on surface) | 2 | R | State: |
| | | | Maintains grip only with no traction | 1 | | |
| | | | No attempt to maintain grasp | 0 | | |
| 4 | Supine head midline | Visual stimulation is given with toy. If head is maintained in midline for 5 | Rotates from maximum rotation to midline | 4 | L>R | Best side: |
| Head in midline with visual | | seconds: Place head in maximum available rotation and provide visual | Turns head part way back to midline | 3 | | |
| stimulation* | | stimulation to encourage midline | Maintains midline for 5 or more seconds | 2 | R>L | State: |
| | | | Maintains midline, less than 5 seconds | 1 | K/L | |
| | | | Head falls to side, no attempts to regain midline | 0 | | |

| Time of eva | luation: | | (AM/PM) Hours off BiPAP at testing: | | | <u>(h)</u> |
|---|---|---|---|---|---|---|
| Item | Position | Test Procedure | Graded Response | | Score | |
| 5 | Supine, no diaper | Hips flexed and adducted Feet hip width | Keeps knee off surface of bed >5 sec or lifts foot off surface | 4 | L | Best side: |
| Hip adductors | | apart and thighs parallel, knees slightly apart | Keeps knees off surface of bed 1-5 sec | 2 | | State: |
| | | | No attempt to maintain knees off surface | 0 | R | State. |
| 6 | Supine (arms at side) Keep side tested | 1. Holding infant's lower thigh, flex hip and knee and adduct across midline | When traction is applied at the end of the maneuver, rolls to prone with lateral head righting | 4 | To R | Best side: |
| Rolling: elicited from legs* | up roll away from the Side<br>tested | bringing pelvis vertical maintain traction and <i>pause in this position</i> . <b>2.</b> If infant rolls to side apply traction at | Rolls through side lying into prone without lateral head righting, clears weight-bearing arm to complete roll | 3 | | |
| | | a 45° diagonal to body and pause to<br>allow infant to attempt to de-rotate body | Pelvis, trunk and arm lift from support surface, head turns and rolls onto side, arm comes thru to front of body | 2 | To L | State: |
| | | Pelvis and trunk lift from support surface and head turns to side. Arm remains behind trunk | 1 | TOL | | |
| | | | Pelvis lifted passively off support surface. | 0 | | |
| 7 Rolling: side tested up roll away from the Side tested | | | Rolls to prone with lateral head righting | 4 | | |
| | Hold infant at the elbow move toward opposite shoulder maintain traction on limb and <i>pause with the shoulders vertical</i> allow infant to de-rotate | Rolls into prone without lateral head righting; must clear weight-bearing arm completely to finish roll | 3 | To R | Best side: | |
| | | Rolls onto side, leg comes thru and adducts, bringing the pelvis vertical | 2 | | | |
| arms* | side tested up foll away from | 2. if the pelvis achieves vertical continue to provide traction | Head turns to side and shoulder and trunk lift from surface | 1 | To L | State: |
| | | continue to provide traction | Head turns to side; body remains limp or shoulder lifts passively | 0 | | State. |
| | | | Clears hand from surface with antigravity arm movement | 4 | L | |
| <b>8</b> Shoulder and | Side-lying with upper arm at 30° of shoulder extension | Prompt reach for a toy presented at | Able to flex shoulder to 45 degrees, without antigravity arm movement | 3 | L | Best side: |
| elbow flexion | and elbow flexion and supported on body | arm's length at shoulder level (may provide stimulation and <i>observe</i> | Flexes elbow after arm comes off body | 2 | | |
| And horizontal abduction | (restrain lower arm if needed) | spontaneous movement) | Able to get arm off body | 1 | R | State: |
| | | | No attempt | 0 | K | State. |
| | | | Abducts or flexes shoulder to 60 degrees | 4 | | Dant side. |
| 9 | Sitting in lap or on mat with | Present stimulus at midline and at | Abducts or flexes shoulder to 30 degrees | 3 | L | Best side: |
| Shoulder flexion | head and trunk support (20° | shoulder level at arm's length (may provide stimulation and <i>observe</i> | Any shoulder flexion or abduction | 2 | | |
| & Elbow flexion | recline) | spontaneous movement) | Flexes elbow only | 1 | R | G4-4 |
| | | | No attempt to lift arm | 0 | | State: |

AveXis, Inc.

| Time of eva | luation: | | (AM/PM) Hours off BiPAP at testing: | | | <u>(h)</u> |
|---|---|---|---|---|---|---|
| Test Procedure | Graded Response | | Score | | | |
| | | | Extends knee to >45 degrees | 4 | L | Best side: |
| 10 | | Tickle plantar surface of foot or | Extends knee 15 to 45 degrees | 2 | L | Dest side. |
| - | | | Any visible knee extension | 1 | | |
| | | | No visible knee extension | 0 | R | State: |
| | | | Hip flexion or knee flexion >30° | 4 | | |
| 11 | | | Any hip flexion or knee flexion | 3 | L | Best side: |
| | Support at the abdomen with | Stroke the foot or pinch the toe | Ankle dorsiflexion only | 2 | | |
| foot dorsiflexion | $\mathcal{E}$ | | No active hip, knee or ankle motion | 1 | R | State: |
| | | | Hip flexion or knee flexion >30° | 0 | | |
| | | | Attains head upright from flexion and turns head side to side | 4 | | |
| | 1 11 14 1 | Place the infant in ring sit with head | Maintains head upright for >15 sec (for bobbing head control score a 2) | 3 | L | Best side: |
| | | shoulders (front and back) (may delay | Maintains head in midline for >5 sec. with the head tipped in up to 30° of forward flexion or extension | 2 | | |
| Head control | | | Actively lifts or rotates head twice from flexion within 15 seconds (do not credit if movement is in time with breathing) | obbing head control score a 2) 3 L Best th the head tipped in up to 30° 2 flexion within 15 seconds (do ime with breathing) 1 R Standards dhangs 0 | State: | |
| | | | No response, head hangs | 0 | | |
| 13 | | Traction responses pull to sit extend | Flexes elbow | 4 | L | Best side: |
| | Supine | arms at 45 degree angle, to point of | Visible biceps contraction without elbow flexion | 2 | | State: |
| 14 | | nearly fitting nead off surface | No visible contraction | 0 | R | State. |
| 14 | | Traction response: hold in neutral proximal | Lifts head off bed | 4 | | Score: |
| Neck Flexion<br>Score with item | Supine | to wrist and shoulder at 45°, to point of | Visible muscle contraction of SCM | 2 | | State: |
| 13 | | nearly lifting head off surface | No muscle contraction | 0 | | State. |
| 15 | Ventral suspension: Prone, | Ctale demands from male to a Til | Extends head to horizontal plane or above | 4 | | Score: |
| Head/Neck<br>Extension | held in one hand upper | Stoke along spine from neck to sacrum. The coronal axis of the head when parallel to the bed surface = 0 degrees (horizontal) | Extends head partially, but not to horizontal | 2 | | State: |
| (Landau) | abdomen | ocu surrace – o uegrees (norizonităt) | No head extension | 0 | | State. |

Investigational Product: AVXS-101

Protocol Number: AVXS-101-CL-101 Version 14.0 / 21 Apr 2016

| Time of eva | luation: | | (AM/PM) | Hours off BiPAP at testing | g: | | <u>(</u> h |
|---|---|---|---|---|---|---|---|
| Item | Position | Test Procedure | | Graded Response | | Score | |
| 16 | | Stroke Right then Left throacoluml | har | Twists pelvis towards stimulus off axis | 4 | L | Best side: |
| Spinal | Ventral suspension: Prone,<br>held in one hand upper | paraspinals or tickle abdomen or foot of | or tilt in | Visible paraspinal muscle contraction | 2 | | |
| Incurvation<br>(Galant) | abdomen | infants with For infant over 10 kg kne-<br>head may touch | es and | No response | 0 | | State: |
| Total score, l | pest score on each side fo | or each item (maximum 64 | points): | | 1 | - 1 | |
| Comments: | | | | | | | |
| * Adapted from<br>Contractures : | n the Test of Infant Motor Pe | erformance, Campbell, SK; et al | | | nd . 1 1004) | | |
| □ None | | State 1 Deep si | | natal Behavioral Assessment Scale, 2 <sup>1</sup><br>State | | | |
| L R R Kne | e flexion | • | y or semi-dozing | State | | hright look | |
| L □ R □ Ank | le plantar flexion egrees knee extended) | • | pen, considerable acti | | - | origin rook | |
| L - R - Hip : | adductor L $\square$ | $R \square$ ITB contracture | | | | | |
| (Note if leg can | not abduct and ext. rot. to co | ontact surface in supine) | | Testing en | vironment: | | |
| L □ R □ Show | ılder protraction | Ideally test | first thing in the AM | or same time of day about 1 hour after | r feeding | | |
| L □ R □ Elbo | w flexion | Test on a fi | irm padded mat | | | | |
| L □ R □ Necl | k rotation | Diaper /one | esie only unless the in | fant is cold | | | |
| L □ R □ Necl | k lateral flexion | Te | est with toys | | | | |
| □ Plagiocephal | У | M | ay use pacifier only if | needed to maintain state 4 or 5 (see d | efinition). | | |
| □ Fixed spinal | | | | t test) if patient could not be tested DO | | ) | |
| SIGNATURE | <u> </u> | | | <br>DATE | | | |

# APPENDIX 4 BAYLEY SCALE OF INFANT DEVELOPMENT VERSION 3: GROSS AND FINE MOTOR SKILLS SUBPARTS AND SPEECH AND COGNITION SUBPARTS







| | C Item | Materials | Score Criteria and Comments | 200 | re |
|---|---|---|---|---|---|
| | 35. Coins in Slot | Bank<br>5 small coins<br>(pennies, nickels,<br>and/or dimes) | Score: Child places at least three coins into slot. | 1 | 0 |
| | 36. Connecting<br>Blocks: Apart | Connecting<br>block set | Score: Child takes all the blocks apart. | 1 | 0 |
| 28<br>34<br><u>37</u><br>48 | 37. Grasp Series:<br>Intermediate<br>(Tripod) Grasp | Crayon or pencil<br>Sheet of<br>blank unlined<br>white paper | Score: Child grasps crayon or pencil using a static tripod (thumb and two fingers) or quadrupod (thumb and three fingers) grasp while making a mark on the paper. | 1 | - |
| 31 D | 38. Block Stacking<br>Series: | 12 blocks | Trials: 3 Score: Child stacks at least slx blocks. Number of blocks in tallest tower: | | |
| 54 | 6 Blocks | | | 1 | ( |
| | 39. Uses Hand to<br>Hold Paper<br>in Place | Crayon or pencil<br>Sheet of<br>blank unlined<br>white paper | Score: Child holds paper in place with one hand while he or she scribbles or draws with the other. | 1 | |
| 32<br>40<br>41<br>43 | 40. Imitates Stroke<br>Series:<br>Horizontal | 2 crayons<br>Sheet of<br>blank unlined<br>white paper | Score: Child's horizontal stroke is within approximately 30° of your horizontal line. | 1 | 1 |
| 32<br>40<br>41<br>43 | 41. Imitates Stroke<br>Series:<br>Vertical | 2 crayons<br>Sheet of<br>blank unlined<br>white paper | Scare: Child's vertical stroke is within approximately 30° of your vertical line. | 1 | |
| | 42. Connecting<br>Blocks: Together | Connecting block set | Score: Child puts all the blocks together. At least two connector knobs on each block should be correctly aligned and secured to another block. | 1 | |
| 32<br>40<br>41 | 43. imitates Stroke<br>Series:<br>Circular | 2 crayons<br>Sheet of<br>blank unlined<br>white paper | Score: Child produces a mostly curved shape. | 1 | |
| | 44. Builds Train<br>of Blocks | 10 blocks | Score: Child places at least four blocks in a row. | 1 | |
| | 45. Strings 3 Blocks | Shoelace<br>3 blocks<br>with holes | Score: Child strings at least three blocks on shoelace. | 1 | |



| | 81 | tem | Materials | Score Criteria and Comments | Sco | H |
|---|---|---|---|---|---|---|
| | 10. | Holds Head<br>in Midline | Object of interest Stopwatch 5 seconds | Score: Child holds head in midline for at least 5 seconds. | 1 | ( |
| | | Upright While | None | Score: Child holds head erect and steady without support while being moved. | 1 | |
| 12<br>17<br>18<br>18<br>19<br>12<br>12<br>17 | 12. | | Object of interest | Score: Child maintains raised head at least 45" from exam surface for at least 2 seconds. | - | |
| | | | | If child holds head at 90°, record elapsed times | 1 | |
| | 13. | Rights Head | None | Score: Child keeps head balanced and in same plane as body or child overcompensates by tilting head toward the vertical plane. | 1 | |
| | | | | Score: Child actively turns from both sides to his or her back. | | |
| | 14. | Rolls From<br>Side to Back | None | Score: Child actively with their book sides to the street | 1 | |
| | 15. | While Prone | Object of interest | Score: Child elevates head and upper trunk by pushing up on elbows or forearms. | 1 | |
| 21 | Series:<br>Elbows and<br>Forearms | | | | | |
| 16 | Elbows and<br>Forearms 16. Sits With Support<br>Series: | ort Stopwatch | Score: Child tenses muscles in an effort to maintain sitting position. | | | |
| 19 | | Briefly | X | Elapsed time: | 1 | |
| 12 | 17. | While Prone Series: Elbows and Forearms 16. Sits With Support Series: Briefly 17. Controls Head While Prone Series: | Object of | Score: Child maintains head at least 90° from exam surface for at least 5 seconds. | | |
| 17 | | | Stopwatch 5 seconds | et least 3 seconds. | 1 | |
| 15 | 15. Elevates Trunk While Prone Series: Elbows and Forearms 16. Sits With Support Series: Briefly 17. Controls Head While Prone Series: 90° 18. Elevates Trunk While Prone Series: Shifts Weight | Object of | Score: Child shifts weight from one arm to the other. | | | |
| 18<br>21 | | Series: | interest | | | 1 |
| 16 (6) | 19 | Sits With Support | | Score: Child sits with slight support for at least 30 seconds. | | |
| 19 | 1 | | 30 seconds | | 2.4 | 1 |
| | 20 | | Bell or rattle | Score: Child turns from back to both right and left sides. | | 1 |
| | | ************************************** | | | | |
| 15<br>18<br><u>21</u> | 21 | While Prone<br>Series: | Object of<br>Interest | Score: Child supports weight on both hands. | | 1 |



| | Item | Materials | | 300 | ore |
|---|---|---|---|---|---|
| 30<br>31<br><u>34</u> | 34. Crawls Series: | Object of interest | Score: Child makes forward progress of at least 5 feet by crawling on hands and knees. | 1 | 0 |
| 0 | 35. Raises Self to<br>Standing Position | Object of interest | Score: Child raises self to a standing position, using a chair or other convenient object for support. | 1 | 0 |
| | 36. Bounces While<br>Standing | None | Scora: Child bounces up and down at least twice by alternately bending and straightening the knees. | 1 | • |
| 37<br>42<br>43 | 37. Walks Series:<br>With Support | None | Score: Child walks by making coordinated, alternating stepping movements. | 1 | |
| | 34. Crawls Series: Crawl Movement Object of interest Score: Child makes forward progress of at least 5 feet by crawling on hands and knees. Score: Child raises self to a standing position, using a chair or other convenient object for support. Score: Child bounces up and down at least twice by alternately bending and straightening the knees. None Score: Child walks by making coordinated, alternating stepping | 1 | | | |
| Q | | None | Score: Child purposely lowers from a standing to a sitting position in a controlled manner. | 1 | 100.00 |
| | 40. Stands Alone | Mone | Score: Child stands alone for at least 3 seconds after you release his or her hands. | 1 | |
| 46 | | ies: None | Score: Child comes to a standing position, rolling first to a prone or quadruped position, without using any support. | 1 | |
| 37<br>42<br>43 | Annual Control of the | None | Score: Child takes at least three steps without support, even if gait is stiff-legged and wobbly. | 1 | 1 |
| 37<br>42<br>43 | Alone With | None | Score: Child takes at least five steps independently, displaying coordination and balance. | , | |
| | 44. Throws Ball | Small ball | Score: Child purposely throws ball forward. | | 1 |



| | 28 | Item | Materials | Score Criteria and Comments | | ic |
|---|---|---|---|---|---|---|
| | | Shows Visual<br>Preference | Stimulus Book<br>(pp. 7-9)<br>Stopwatch<br>15 seconds<br>per page | Score: Child looks longer at striped pattern on both pages. | 1 | |
| | 12. | Habituates<br>to Object | 2 blocks without<br>holes<br>Stopwatch<br>30 seconds | <b>Score:</b> Child habituates within 30 seconds, displaying decrease in attention and interest. | 1 | |
| | 13. | Prefers Novel<br>Object | Block without<br>hole<br>Small ball<br>Stopwatch<br>15 seconds per<br>presentation | Score: Child looks longer at ball than block in both presentations. | 1 | |
| | 14. | Habituates to<br>Picture (Balloons) | Stimulus Book<br>(p. 11)<br>Stopwatch<br>30 seconds | Score: Child habituates within 30 seconds, displaying decrease in attention and interest. | 1 | |
| | 15. | Prefers Novel<br>Picture (Ball) | Stimulus Book<br>(pp. 13–15)<br>Stopwatch<br>15 seconds<br>per page | Score: Child looks longer at ball than balloons in both presentations. | 1 | |
| (3) | 16. | Explores Object | Rattle or other<br>small object<br>of interest | Score: Child attends to sight, sound, or feel of object by shaking, mouthing, or other activity. | 1 | The second secon |
| | 17. | Carries Object<br>to Mouth | Glitter bracelet<br>or other small<br>object of interest | Score: Child purposely carries object to mouth. | 1 | |
| | 18. | Inspects Own<br>Hand | None | Score: Child visually inspects one or both hands. | 1 | |
| 1 <u>9</u> (F) | 19. | Mirror Image<br>Series:<br>Approaches | Mirror | Score: Chi'd approaches mirror image with head, body, or hands, or purposely touches mirror image. | 1 | |
| 2<br>20 | 20. | Responds to<br>Surroundings<br>Series:<br>Awareness<br>of Novelty | Nene | Score: Child displays awareness of being in novel surroundings (e.g., startles, looks around). | 1 | |
| | 21, | Per sistent Reach | Block without<br>hole or other<br>small object<br>of interest | <b>Score:</b> Child persistently reaches for object, even if he or she fails to obtain it. | 1 | |

| - | € | | Materials | Score Criteria and Comments | Score |
|---|---|---|---|---|---|
| 2 | 22. | Mirror Image<br>Series:<br>Responds<br>Positively | Mirror | Score: Child plays with image by looking and smiling/laughing, patting, banging, reaching playfully, or mouthing. | 1 0 |
| | 23. | Plays With String | Ring with string | Score: Child plays with string by picking it up, chewing it, pulling on it, or manipulating it. | 1 0 |
| | 24. | Bangs in Play | Block without<br>hole, spoon, or<br>other suitable<br>hard object | Score: Child purposely bangs in play at any time during testing. | 1 0 |
| <b>(F)</b> | 25. | Searches for<br>Fallen Object | Squeeze toy | Score: Child looks for fallen toy by looking toward floor. | 1 0 |
| 6 | 26. | Bell Series:<br>Manipulates | Bell | Score: Child manipulates bell while looking at it with interest. | 1 0 |
| 7 3 7 | 27. | Picks Up Block<br>Series:<br>Reaches for<br>Second Block | 3 blocks<br>without holes | Score: Child holds first block and reaches for second block. | 1 0 |
| | 28. | Pulls Cloth to<br>Obtain Object | Washcloth<br>Object of interest | Score: Child pulls washcloth purposely toward him or her to obtain object. | 1 0 |
| | 29. | Pulls String<br>Adaptively | Ring with string | Score: Child picks up string, purposely pulls to secure ring, and grasps ring. | 1 0 |
| | 30. | Retains Both<br>Blocks | 2 blocks<br>without holes | Score: Child holds both blocks simultaneously for at least 3 seconds. | 1 0 |
| 6 | 31. | Bell Series:<br>Rings Purposely | Bell | Score: Child holds bell by handle and purposely rings it. | 1 0 |
| | 32. | Looks at Pictures | Picture Book | Score: Child regards one or more specific pictures with interest or recognition. | 1 0 |
| 27<br>33<br>37 | 33. | Picks Up Block<br>Series:<br>Retains 2 of<br>3 Blocks | 3 blocks<br>without holes | Score: Child retains first two blocks for at least 3 seconds after visually attending to third block. | 1 ( |

| | Si | Item | Materials | Score Criteria and Comments | 5 | co |
|---|---|---|---|---|---|---|
| 0 | 34. | Searches for<br>Missing Objects | 3 blocks<br>without holes<br>Cup with handle | Trials 2 Score: Child looks into empty cup for blocks. | 1 | |
| | 35. | Takes Blocks<br>Out of Cup | 3 blocks<br>without holes<br>Cup with handle<br>Stopwatch | Score: Child takes all three blocks out of cup. | 1 | lin. |
| 36<br>54 | 36. | Block Series<br>1 Block | 9 blocks<br>Cup with handle | Score: Child places at least one block in or over cup, even if he or she does not release it. Number of blocks in cup: | , | |
| 27<br>33<br><u>37</u> | 37. | Picks Up Block<br>Series:<br>3 Blocks | 3 blocks<br>without holes | Score: Child retains first two blocks in one or both hands and attempts to secure third block. | 1 | |
| | 38. | Explores Holes<br>in Pegboard | Pegboard | Score: Child intentionally pokes finger into at least one hole. | .1 | 1 |
| | 39. | Pushes Car | Car | Score: Child intentionally pushes car so that all four wheels stay on table. | 7 | - |
| <b>®</b> | 40. | Finds Hidden<br>Object | Glitter bracelet<br>2 washcloths | Trial: 2 Score: Child finds bracelet by looking first under correct washcloth when hidden on both left and right sides. Trial 1 | 1 | |
| | 41. | Suspends Ring | Ring with string | Score: Child obtains ring and suspends it by string without the ring touching the table. | 1 | 1 |
| | 42. | Removes Pellet | Food pellet<br>Bottle<br>(without lid) | Trials: 3 Score: Child purposely removes pellet from bottle using some form of directed effort. | 1 | - |
| | 43. | Clear Box: Front | Clear box Small object of interest Stopwatch | Score: Child retrieves object through open end of box within 20 seconds. | 1 | ( |
| | 44. | Squeezes Object | Squeeze toy | Score: Child attempts to squeeze toy to make the sound. | 1 | ( |

| - | | Item | Materials | Score Criteria and Comments | Sea | r |
|---|---|---|---|---|---|---|
| (8) | 43. | Finds Hidden<br>Object (Reversed) | Glitter bracelet<br>2 washcloths | Trials: 2 Score: Child finds bracelet by looking first under correct washcloth when hidden on both left and right sides. Trial 1 | 1 | 0 |
| | 46. | Removes Lid<br>From Bottle | Bottle with lid | Score: Child unscrews lid until it comes off. | 1 | 0 |
| | 47. | Pegboard Series:<br>2 Holes | Pegboard<br>6 yellow pegs | Trials: 3 Score: Child places at least one peg two or more times in the same or different hole(s). | | |
| | | | Trials: 3 Score: Child places at least one peg two or more times in the same or different hole(s). Trial 1 Completion time (all 6 pegs): Trial 2 Completion time (all 6 pegs): Trial 3 Completion time (all 6 pegs): Trial 2 Completion time (all 6 pegs): Trial 2 Completion time (all 6 pegs): Trial 3 Completion time (all 6 pegs): Trial 3 Completion time (all 6 pegs): Trial 2 Completion time (all 6 pegs): Trial 2 Completion time (all 6 pegs): Trial 3 Completion time (all 6 pegs | | | |
| | | | | The second secon | 1 | 0 |
| | | | per trial | Trial 3 Completion time (all 6 pegs): | e (all 6 pegs): e (all 6 pegs): e (all 6 pegs): 1 0 ates relational play using him- or herself. 1 1 places at least one piece within 180 seconds. ly (180 seconds): | |
| | 48. | Relational Play | Doll | Score: Child demonstrates relational play using him- or herself. | | _ |
| | | Series:<br>Self | Plastic cups<br>Spoons<br>Small ball<br>Washcloths | | 1 | ( |
| | 49. | Pink Board Series: | Pink board | Score: Child correctly places at least one piece within 180 seconds. | | |
| | | 1 Piece | (square, circle,<br>triangle)<br>Stopwatch | # pieces placed correctly (180 seconds): | 1 | ( |
| | 50. | Finds Hidden<br>Object (Visible | 4.00 | | | |
| | | Displacement) | | Trial 1 | 1 | • |
| | 51. | Blue Board Series: | Blue board | Score: Child correctly places at least one piece within 150 seconds. | | |
| | | 1 Piece | Blue block<br>set (4 round, | Completion time: # of pieces: | | |
| | | | 5 square)<br>Stopwatch | | 1 | C |
| | 52. | Clear Box: Sides | Clear box Small object of interest Stopwatch 20 seconds per side | <b>Score:</b> Child retrieves object through open end of box when presented on both left and right sides. | 1 | 0 |

AveXis, Inc. Investigational Product: AVXS-101

| _ | E I | term | Materials | Score Criteria and Comments | 5 | Sc |
|---|---|---|---|---|---|---|
| 48<br><u>53</u> | | Relational Play<br>Series<br>Others | Doll<br>Bear<br>Plastic cups<br>Spoons<br>Small ball<br>Washcloths<br>Several blocks | Score: Child demonstrates relational play, using objects for how they are intended, with others. | 1 | |
| 36<br><u>54</u> | | Block Series:<br>9 Blocks | 9 blocks<br>Cup with handle | Score: Child places all nine blocks inside cup at one time. # of blocks in cup: | 1 | |
| | 55. | Pegbrard | Pegboard | Trials: 3 Score: Child places all six pegs in pegboard within 70 seconds. | | |
| 47 | | Series: 6 Pegs | 6 yellow pegs | Trial 1 Completion time (all 6 pegs): | + | |
| <u>55</u> | | 3000000000000 | Stopwatch | the state of the s | + | |
| | | | 70 seconds | Trial 2 Completion time (all 6 pegs): | 1 | ı |
| | | | g / v securas | Trial 3 Completion time (all 6 pegs): | | |
| | 0.00 | Pink Board | Pink board | Score: Child correctly places all three pieces within 180 seconds. | | |
| <u>56</u> | | Series:<br>Completes | Red block set<br>(square, circle, | # pieces placed correctly (180 seconds): | | |
| • | | | triangle)<br>Stopwatch<br># 180 seconds | | 1 | |
| | | Uses Pencil to<br>Obtain Object | Pencil<br>Small red duck | Trials: 2 Score: Child uses pencil to attempt to obtain duck. | 1 | |
| 51 | | Blue B¢ ard | Blue board | Score: Child correctly places at least four pieces within 150 seconds. | | |
| <u>58</u><br>66 | | Series<br>4 Pieces | Blue block<br>set (4 round,<br>5 square)<br>Stopwatch | Completion time: # of pieces: | 1 | |
| | 59. / | Attends to Story | Story Book | Score: Child attends to entire story | 1 | |
| 0 | 60. | Rotated Pink | Pink board | Score: Child correctly places all three pieces while board is in | | |
| 9 | | Board | Red block set<br>(square, circle,<br>triangle) | rotated position. | 1 | |
| | | Object Assembly<br>(Ball) | Ball puzzle<br>Stopwatch | Trials: 2 Score: Child correctly assembles object within 90 seconds in either trial. | 1 | |
| | - | Completes<br>Pegboard: | <ul> <li>90 seconds</li> <li>Pegboard</li> <li>6 yellow pegs</li> </ul> | Score: Child places all six pegs in pegboard within 25 seconds. | | |
| | | 25 Seconds | Stopwatch 25 seconds | | 1 | |

| | Sai | Item | Materials | Score Criteria and Comments | Sco | iL.S |
|---|---|---|---|---|---|---|
| Ø | 63. | Object Assembly<br>(Ice Cream Cone) | Ice cream cone<br>puzzle<br>Stopwatch<br>• 90 seconds | Trials: 2 Score: Child correctly assembles object within 90 seconds in either trial. | 1 | 0 |
| | 64. | Matches Pictures | Stimulus Book<br>(pp. 17–23) | Score: Child correctly identifies matching picture on at least three pages. Airplane Tricycle Tree Telephone | 1 | 0 |
| | 65. | Representational<br>Play | Plastic cups<br>Spoon<br>Doll<br>Washcloths<br>Block<br>Other objects<br>of interest | Score: Child takes an object and pretends it is something else. | 1 | C |
| | 66. | Blue Board<br>Series:<br>Completes<br>(75 Seconds) | Blue board Blue block set (4 round, 5 square) Stopwatch 75 seconds | Score: Child correctly places all nine pieces within 75 seconds. | 1 | |
| <b>(9)</b> | 67. | Imitates a Two-<br>Step Action | Small yellow<br>duck<br>Spoon | Trials: 3 Score: Child correctly imitates both steps. | 1 | ( |
| | 68. | Matches 3 Colors | Stimulus Book<br>(p. 25)<br>Red, yellow, blue,<br>and green disks | Score: Child places yellow, blue, and green disks on or near matching crayons in Stimulus Book, or points to matching crayons. Yellow Blue Green | 1 | 0 |
| | 69. | Imaginary Play | Plastic cups<br>Spoon<br>Doll<br>Bear<br>Washcloths<br>Small ball<br>Other objects<br>of interest | Score: Child uses imaginary objects in play. | 1 | ( |
| | 70. | Understands<br>Concept of One | 3 blocks<br>without holes<br>Stopwatch<br>5 seconds | Score: Child hands you only one block within 5 seconds. | 1 | ( |
| | 71. | Multischeme<br>Combination Play | Plastic cups | Score: Child demonstrates multischeme combination play involving at least two steps. | 1 | ( |

AveXis, Inc. Investigational Product: AVXS-101

| Score: Child correctly identifies both blue ducks. | SI | - Item | Materials | Score Criteria and Comments |
|---|---|---|---|---|
| 273. Concept Grouping: Size Sig and little ducks (red and yellow) 274. Compares Masses 2 big blue ducks Score: Child correctly identifies both little ducks and both big ducks. 275. Matches Size Big red duck Sig blue duck Little yellow duck Little yellow duck Little yellow duck Little yellow duck Score: Child correctly identifies big blue duck Little yellow duck Little yellow duck Score: Child correctly identifies salf and donkey. 276. Discriminates Stimulus Book (pp. 27-37) Simple Pattern Big and little ducks Score: Child correctly identifies salf and donkey. 277. Simple Pattern Big and little ducks Score: Child correctly identifies big yellow duck. 278. Sorts Pegs 4 red pegs 4 yellow pegs 3 plastic cups Score: Child sorts pegs by color, placing them in appropriate cups or in separate piles. 279. Counts Concison Stimulus Book (pp. 39-43) Score: Child assigns only one number to each block when counting. Child must count to at least 3 in proper sequence. 380. Discriminates Stimulus Book (pp. 39-43) Score: Child identifies correctly-ized object for at least two of three pages. 381. Identifies 3 (pp. 45-61) Box lid | 72 | | | Score: Child correctly identifies both blue ducks. |
| Grouping: Size ducks feed and yellow) | | Grouping: Color | | |
| 2 big blue duck Trials: 2 Score: Child correctly identifies heavy duck when placed in both left and right hands. 75. Matches Size Big red duck Big blue duck Little yellow duck Little yellow duck Little yellow duck Score: Child correctly identifies big blue duck Score: Child correctly identifies calf and donkey. 76. Discriminates Stimulus Book (pp. 27-37) Simple Pattern Big and little ducks Score: Child correctly identifies big yellow duck, 77. Simple Pattern Big and little ducks Score: Child correctly identifies big yellow duck, 78. Sorts Pegs 4 red pegs 4 yellow pegs 4 blue pegs 3 plastic cups 79. Counts (One-to-One Correspondence) S blocks Score: Child sorts pegs by color, placing them in appropriate cups or in separate piles. 80. Discriminates Stimulus Book (pp. 39-43) Score: Child dentifies correctly-sized object for at least two of three pages. 81. Identifies 3 Incomplete Pictures Stimulus Book (pp. 45-61) Face Cat Flower 82. Object Assembly (Dog) Dog puzzle Stimulus Book Stores Stimulus Book (pp. 45-61) Face Cat Flower 83. Discriminates Stimulus Book Sti | 73 | | | Score: Child correctly identifies both little ducks and both big ducks. |
| Masses Big red duck Big blue duck Little yellow duck Score: Child correctly identifies big blue duck Little yellow duck Score: Child correctly identifies calf and donkey. | | Grouping, Size | | |
| Big blue duck Little yellow duck | 74. | | 2 big blue ducks | Trials: 2 Score: Child correctly identifies heavy duck when placed in both left and right hands. |
| Big blue duck Little yellow duck Little yellow duck Score: Child correctly identifies calf and donkey. | | | | |
| Little yellow duck | 75. | Matches Size | | Score: Child correctly identifies big blue duck |
| Pictures (pp. 27-37) Pictures (pp. 27-37) | | | | |
| 77. Simple Pattern Big and little ducks Score: Child correctly identifies big yellow duck. Score: Child correctly identifies big yellow duck. Score: Child sorts pegs by color, placing them in appropriate cups or in separate piles. Score: Child assigns only one number to each block when counting. Child must count to at least 3 in proper sequence. Score: Child dentifies correctly-sized object for at least two of three pages. Score: Child identifies correctly-sized object for at least two of three pages. Box lid | 76. | | | Score: Child correctly identifies calf and donkey. |
| 78. Sorts Pegs by Color 4 red pegs 4 yellow pegs 4 blue pegs 3 plastic cups 79. Counts (One-to-One Correspondence) 80. Discriminates Sizes Stimulus Book (pp. 39–43) 81. Identifies 3 Incomplete Pictures Stimulus Book (pp. 45–61) Dog puzzle Stopwatch 9 0 seconds Stimulus Book Ratherer Stimulus Book (pp. 45–61) Dog puzzle Stopwatch 9 0 seconds Score: Child correctly identifies image when presented with first or second page of the series. Trials: 2 Score: Child correctly assembles object within 90 seconds in either trial. Score: Child correctly identifies image when presented with first or second page of the series. Face Cat Trials: 2 Score: Child correctly assembles object within 90 seconds in either trial. | | Tan cooks | | |
| Score: Child assigns only one number to each block when counting. Counts (One-to-One Correspondence) Stimulus Book (pp. 39–43) | 77. | Simple Pattern | | Score: Child correctly identifies big yellow duck, |
| Score: Child assigns only one number to each block when counting. Counts (One-to-One Correspondence) Stimulus Book (pp. 39–43) | | | | |
| 79. Counts (One-to-One Correspondence) 80. Discriminates Sizes 81. Identifies 3 Incomplete Pictures 82. Object Assembly (Dog) 83. Discriminates 84. Discriminates 85. Discriminates 86. Discriminates 87. Stimulus Book (pp. 45-61) 88. Stimulus Book (pp. 45-61) 88. Stimulus Book (pp. 45-61) 88. Stimulus Book (pp. 45-61) 88. Stimulus Book (pp. 45-61) 88. Object Assembly (Dog) 88. Discriminates 88. Stimulus Book 88. Discriminates 88. Discriminates 88. Discriminates 88. Stimulus Book 89. Stimulus Book 89. Score: Child correctly identifies out of-place object for all three pages. | 78. | | 4 yellow pegs | Score: Child sorts pegs by color, placing them in appropriate cups or in separate piles. |
| Child must count to at least 3 in proper sequence. Child must count to at least 3 in proper sequence. Child must count to at least 3 in proper sequence. Child must count to at least 3 in proper sequence. Score: Child dentifies correctly-sized object for at least two of three pages. Box lid | | | | |
| 80. Discriminates Stimulus Book (pp. 39–43) 81. Identifies 3 Incomplete Pictures Stimulus Book (pp. 45–61) Score: For all three series, child correctly identifies image when presented with first or second page of the series. □ Face □ Cat □ Flower Trials: 2 Score: Child correctly assembles object within 90 seconds in either trial. Score: Child correctly identifies out of-place object for all three pages. Score: Child correctly identifies out of-place object for all three pages. | 79. | (One-to-One | 5 blocks | Score: Child assigns only one number to each block when counting. Child must count to at least 3 in proper sequence. |
| 81. Identifies 3 Incomplete Pictures Stimulus Book (pp. 45–61) Box lid □ Bowl □ Shoe Score: For all three series, child correctly identifies image when presented with first or second page of the series. □ Face □ Cat □ Flower Trials: 2 Score: Child correctly assembles object within 90 seconds in either trial. Score: Child correctly identifies out of-place object for all three pages. | | Correspondence) | | |
| 81. Identifies 3 Stimulus Book (pp. 45–61) Score: For all three series, child correctly identifies image when presented with first or second page of the series. | 80. | | | |
| Incomplete Pictures | | 1 | (Pp. 11. 10) | □ Box lid □ Sowl □ Shoe |
| Pictures □ Face □ Cat □ Flower Plower Plo | 81. | | | Score: For all three series, child correctly identifies image when presented |
| (Dog) Stopwatch 90 seconds 83. Discriminates Stimulus Book Patterns (no. 63 67) Store: Child correctly identifies out of-place object for all three pages. | | | (pp. 43-61) | |
| (Dog) Stopwatch 90 seconds Store: Ch'ld correct y identifes out of-place object for all three pages. | | | | |
| 83. Discriminates Stimulus Book Patters: (no. 63. 67) Score: Ch'ld correctly identifies out of-place object for all three pages. | 82. | | | |
| Patterns (no. 62, 67) | | | 1000 000 00 | |
| Patterns (pp. 63-67) Square Triangle E | 83. | | VALUE OF THE PROPERTY OF THE PARTY OF THE PA | Score: Child correctly identifies out of-place object for all three pages. |
| | | ratterns | (pp. 63-67) | □ Square □ Triangle □ E |

| rds for the first | | | Score Criteria | Materials | Item | w |
|---|---|---|---|---|---|---|
| | correct pairs of ca | rrectly identifies the | Score: Child co<br>two objects. | Memory Cards | Spatial Memory | 84. |
| 1 0 | □ Cars | ☐ Flowers | Tops | | | |
| | both parts. | errectly responds to | Score: Child co | 10 blocks | Counts | 85. |
| 1 0 | | | | | (Cardinality) | |
| | h questions. | rrectly answers bot | Score: Child co | 5 blocks | Number | 86. |
| 1 0 | | | | | Constancy | |
| , in proper order | h entire lacing card<br>ound side of card. | ces shoelace throug<br>g holes or lacing an | Score: Child la<br>without skippin | Lacing card<br>Shoelace | Laces Card | 87. |
| don't belong. | THE RESERVE OF THE PARTY OF THE | orrectly identifies all | | Stimulus Book | Classifies Objects | 88. |
| 1 0 | □ Train | □ Lamp | ☐ Banana | (pp. 69-73) | | |
| ions. | all four administrat | errectly responds to | Score: Child c | 9 blocks | Understands | 89. |
| ☐ Fourth | ☐ Third | ☐ Second | ☐ First | 1 red disc | Concept of More | |
| quences. | ast four number se | rrectly repeats at le | Score: Child co | None | Repeats Number | 90. |
| | | A. S. A. S. A. S. A. S. A. S. S. A. S. | ☐ A: 4-2-5 | 10.0000 | Sequences | |
| | | | □ B: 3-1-4-2 | | | |
| | | | □ C: 7-9-1-3 | | | |
| 1 0 | | | □ D: 5-3-7-1- | | | |
| | | -4 | □ E: 8-1-9-6 | | | |
| ree patterns | pegboard for all th | aces correct pegs in | | Pegboard | Completes | 91. |
| | | | Pattern 1 🗆 R- | Red, blue, and<br>yellow pegs | Patterns | |
| 1 0 | | | Pattern 2 C Y- | Jenott pegs | | |
| | | [-0-1- <b>1-D</b> | Pattern 3 🗆 Y- | | | |
| | Total R | | | | 77 | |

Protocol Number: AVXS-101-CL-101 Version 14.0 / 21 Apr 2016

# APPENDIX 5 GROSS MOTOR SKILLS CHECKLIST

| Subj | ect: | Date: | Evaluato | OC. | | |
|---|---|---|---|---|---|---|
| Item Description 1. Hands to midline in supine | Image | Able to<br>Perform<br>Yes | | s in | Yes D | N |
| Holds<br>head<br>upright<br>while<br>carried | | Yes | No 7. Sits w | | Yes | N |
| 3. Lifts<br>head in<br>prone | 30- | Yes | No 8. Rolls from back stome | to -000 | Yes | N |
| 4. Rolls<br>from<br>side to<br>back | | Ye | 9. Rolls<br>from<br>stoms<br>to ba | ach D | Yes | N |
| 5. Rolls<br>from<br>back to<br>side | | Ye. | No 10. Sits without support | | Yes | N |

AveXis, Inc. Investigational Product: AVXS-101

| Item<br>Description | Image | Able<br>Perfor | | 14. Cruises<br>at<br>support | Yes | No |
|---|---|---|---|---|---|---|
| 11. Sits without support and plays | | Yes | No | surface | | |
| 12. Holds<br>hands<br>and<br>knees<br>position | | Yes | No | 15. Walks<br>with<br>support | Yes | No |
| 13. Pulls to<br>Stand | in in | Yes | No | 16.<br>Takes<br>independent<br>steps | Yes | No |